# Implementation and Evaluation of the Pathway Platform: A Digitally Enabled Care Pathway to Improve Depression Key Performance Indicators and Patient Outcomes in Primary Care Clinics

#### **Principal Investigator:**

Dr. David Kemp
Behavioral Health Director
Advocate Health Care
David.Kemp@aah.org

#### **Collaborators:**

Takeda Pharmaceuticals USA, Inc.

Lundbeck LLC, USA

Mobile App for Patients and Care Team Interface Powered by Fora Health, a Ctrl Group Ltd Product

### **TABLE OF CONTENTS**

| S | UMMA | ARY | 4 |
|---|---|---|---|
| | Study | Title | 4 |
| | Object | tives | 4 |
| | Design | n and Outcomes | 4 |
| | Sampl | e Size and Population | 4 |
| L | IST O | F ABBREVIATIONS | 7 |
| 1 | ST | UDY OBJECTIVES | 8 |
| | 1.1 | Primary Objective | 8 |
| | 1.2 | Secondary Objectives | 8 |
| 2. | . BA | ACKGROUND AND RATIONALE | 8 |
| | 2.1 | Background | 8 |
| | 2.2 | Study Rationale | |
| 3. | . ST | TUDY DESIGN | 10 |
| | 3.1 | Performance among participating clinics post-implementation | 11 |
| | 3.2 | Retrospective Assessment: pre-implementation performance at the clinic level Pathway Platform implementation) | el (before |
| 4. | . SE | LECTION AND ENROLLMENT OF PARTICIPANTS | |
| | 4.1 | Inclusion | 12 |
| | 4.2 | Exclusion | |
| | 4.3 | Study Enrollment Procedures | |
| | 4.4 | Pathway Platform | |
| | 4.4. | | |
| | 4.4. | 2 Electronic Medical Record integration | 15 |
| | 4.4. | 3 Educational Scaffolding | 15 |
| | 4.5 | Study Duration | 16 |
| 5. | . ST | UDY PROCEDURES | 16 |
| | 5.1 | Schedule of events | 16 |
| | 5.2 | Description of study evaluations | 18 |
| 6. | . SA | FETY ASSESSMENTS | 18 |
| | 6.1 | Adverse Events Related to the Pathway Platform | |
| | 6.2 | Change in Participant Suicidal Ideation | |
| 7. | . IN | TERVENTION DISCONTINUATION | |

| 8. | ST | FATISTICAL CONSIDERATIONS | 20 |
|-----|-------|-------------------------------------------------------|----|
| 8 | .1 | General Design and Hypothesis | 20 |
| 8 | .2 | Sample size and randomization | 20 |
| 8 | .3 | Outcomes | 21 |
| | 8.3.1 | .1 Primary outcome | 21 |
| | 8.3.2 | .2 Secondary outcome | 21 |
| | 8.3.3 | .3 Exploratory outcomes | 22 |
| | 8.3.4 | .4 Patient and provider in-depth interviews | 23 |
| | 8.3.5 | .5 System level performance | 24 |
| 8 | .4 | Data analysis | 24 |
| 9. | PA | ARTICIPANT RIGHTS AND CONFIDENTIALITY | 25 |
| 9 | .1 | Institutional Review Board (IRB) Review | 25 |
| 9 | .2 | Informed Consent Forms | 25 |
| 9. | .3 | Participant Confidentiality | 25 |
| 9 | .4 | Study Discontinuation | 26 |
| 10. | | AKEDA MARKETED PRODUCT ADVERSE EVENT R<br>EQUIREMENTS | |
| 1 | 0.1 | Special Situation Reports and Product Quality Issues | 26 |
| 1 | 0.2 | Procedures | 27 |
| 11. | PU. | UBLICATION OF RESEARCH FINDINGS | 27 |
| 12 | DF | FEFDENCES | 27 |

#### **SUMMARY**

#### **Study Title**

Implementation and Evaluation of a Digitally Enabled Care Pathway to Improve Depression Key Performance Indicators and Patient Outcomes in Primary Care.

#### **Objectives**

The primary objective of this study is to determine whether implementing the Pathway Platform in primary care improves adherence to measurement-based care practices.

Secondary objectives include determining whether implementing the Pathway Platform improves additional clinical process measures and depression response and remission outcomes.

#### **Design and Outcomes**

A pre- and post- study design is utilized to assess the impact of implementing the Pathway Platform in the primary care setting. Up to 20 primary care sites will be identified to participate in the study. Care team members involved in depression management will receive education on evidence-based clinical practices for depression care, such as measurement-based care practices and shareddecision making. Clinics with behavioral resources will also receive additional education on behavioral health integration. Training on how to onboard patients to use the Pathway Platform and utilize electronic medical records to view data collected in the Pathway Platform will also be provided. Study outcomes identified in this protocol will be assessed among 200 patients who will be enrolled in the Pathway Platform (post-implementation cohort). Outcomes will also be assessed in another 200 patients from the same participating clinics prior to study implementation (preimplementation cohort). Implementation success will be evaluated by comparing study outcomes among the two cohorts with a total sample size of 400 patients (of which 200 will receive the intervention and 200 will not). The primary outcome is PHQ-9 utilization over six months and will be compared between the pre- and post- implementation cohorts. Additional process measures will be compared, including shared-decision making, medication adjustments, referrals to behavioral health, primary care follow-up post hospitalizations, and remission and response. Data collected in the Pathway Platform will also be evaluated to explore pre-defined patient outcomes. Additional outcomes will be explored in data captured from patients who continue to use the app beyond the initial 6 month study period.

#### Sample Size and Population

The study will take place in up 20 primary care clinics within Advocate Aurora Health Care that are representative of different geographic locations, patient populations, and care models for

depression management, including behavioral health integration models.

The Pathway Platform consists of a mobile app for patients and a care team interface that can be accessed through Epic. We intend to enroll 200 patients who meet the eligibility criteria for this study and agree to download the Pathway Platform. An additional 200 patients will be identified from the same participating clinics to form the pre-implementation cohort. These are patients who visited the participating clinics at least 6 months prior to study implementation; they will not be actively enrolled into the study and their data will be collected retrospectively through chart reviews and electronic data pulls.



#### LIST OF ABBREVIATIONS

AE Adverse Event

APA American Psychiatric Association

APPS Mobile Health Applications

ASEX Arizona Sexual Experience Scale

CCM Collaborative Care Model

DSST Digit Symbol Substitution Test

ED Emergency Department
EMR Electronic Medical Record
GAD Generalized Anxiety Disorder

GAS Goal Attainment Scale

GAD Generalized Anxiety Disorder IRB Institutional Review Board

IOR Interquartile Range

MBC Measurement Based Care
MDD Major Depressive Disorder
PAM-13 Patient Activation Measure

PDO-D5 Perceived Deficits Questionnaire- Depression

PHQ-2 Patient Health Questionnaire-2

PHO-9 Patient Health Questionnaire Depression

PROMIS Patient-Reported Outcomes Measurement Information System

PSD-6 PROMIS Sleep Disturbance 6a PTSD Post-Traumatic Stress Disorder

SAE Serious Adverse Event SD Standard Deviation

SDM Shared-Decision Making Model

SSR Special Situation Report

WSAS Work and Social Adjustment Scale

WHO-5 World Heart Organization- Five Well Being Index

#### 1 STUDY OBJECTIVES

#### 1.1 Primary Objective

The primary objective of this study is to determine whether implementing the Pathway Platform in primary care improves adherence to measurement-based care practices. We hypothesize improved clinical processes in measurement-based care, measured by PHQ-9 utilization among patients attending clinics post-implementation compared to those attending clinics pre-implementation.

#### 1.2 Secondary Objectives

Secondary objectives include determining whether implementing the Pathway Platform improves additional clinical process measures and MDD response and remission outcomes. Patient outcomes and Pathway Platform utilization will be explored among patients using the Pathway Platform.

#### 2. BACKGROUND AND RATIONALE

#### 2.1 Background

Health-related technology solutions that utilize mobile phones, known as mobile health applications (apps), have the potential to expand health interventions beyond the traditional face-to-face patient visit. For the healthcare provider, mobile apps can offer low cost and easily scalable interventions to monitor and improve services to patient populations that are difficult to retain in treatment and may promote better health. Uptake of health-related mobile apps has increased in recent years as technology barriers such as access, knowledge, and product usability have improved, reducing obstacles for 'digitally excluded' subpopulations (e.g., poor, rural, and older). Consensus exists that the availability of a mobile app for depression management that is user friendly and aligns with busy office practice would likely be adopted by end users. A Patients with depression and their treating provider may benefit from the use of a mobile health app to assist in disease management.

American Psychiatric Association (APA) clinical guidelines recommend measurement-based care (MBC) in treating depression, defined as a psychiatric evaluation including quantitative measures of symptoms, level of functioning, and quality of life. APA guidelines cite several studies that have shown benefits in using quantitative measures during an initial screening and also for monitoring depression throughout treatment. A mobile app may promote MBC by allowing patients to remotely answer quantitative instruments, such as the PHQ-9, which can be uploaded into their electronic medical records (EMR) for in office visits and physician monitoring. A study

by Torous et al. found that while in person paper scores and app scores were strongly correlated (r=.84), PHQ-9 app scores were consistently higher over a 30 days period.<sup>6</sup> An overall conclusion of this study was that collecting PHQ-9's through a mobile app may be more sensitive than the traditional PHQ-9.<sup>6</sup> Increased consultation times are often cited as a barrier to MBC implementation.<sup>5,7</sup> An app may save time as the physician will only need to review PHQ-9 instead of administering the questions during the visit. Although the validity of the PHQ-9 has been shown in studies, further research is needed to assess its ability to track outcomes of depression therapy over time.<sup>7</sup> This systematic approach to treatment may have positive effects on the patient-physician relationship and enhance shared decision making.<sup>5</sup>

A shared decision-making (SDM) model of interaction can foster patient provider engagement as well as increase patient satisfaction. Several studies have found that individuals suffering from a mental illness want a larger part in the treatment decision making process. A common barrier for SDM is a physician choosing a treatment plan that is not mutually agreed on by both the physician and patient. This can be overcome by increasing education and further clarifying the benefits of a specific treatment plan to align with the patient's values. Incorporating a SDM model may help increase adherence to drug treatment in a primary care setting. Mobile technology can enhance SDM.

A collaborative care model (CCM) that involves behavioral health integration within primary care is another evidence-based practice that enhances depression management. Collaborative care is a systematic approach that improves patient education and integrates mental health professionals or other care extenders, such as nurses, into the primary care clinic to help primary care physicians provide treatment in conformity with evidence-based guidelines.<sup>10</sup> CCM's have been shown to improve outcomes of patients with major depression.<sup>11</sup>

We hypothesize that integrating the Pathway Platform to support measurement- based care and shared decision- making, will improve the clinic workflow, depression management, adherence to medication, patient-provider engagement and improve depression outcomes and care.

#### 2.2 Study Rationale

Major Depressive Disorder (MDD) is a serious public health concern worldwide with ample documentation demonstrating that it is one of the leading contributors to the global burden of disease and is currently the leading cause of disability worldwide. Moreover, the economic burden of MDD is estimated to total \$210.5 billion with approximately 50% of the cost being attributable to impairment in role function. MDD is estimated to total \$210.5 billion with approximately 50% of the cost being attributable to impairment in role function.

A selection of mobile apps has been developed and are available for depression management.

However, many are patient facing only and have not implemented a care team interface. Most of these apps have been assessed for effectiveness in a research setting only and have not been integrated within clinic workflow resulting in lack of adoption by the care team and by healthcare systems.

This study builds on prior work that piloted a mobile App for feasibility and depression management, the *Pathway app*. The first iteration of the Pathway App included patient reported outcomes related to depression, wellbeing, cognitive symptom tracking, medication adherence and side effects. Pilot results confirmed the feasibility of using the Pathway app in patients with depression and showed a trend in patient engagement in the app arm, albeit in a small sample size. The Pathway pilot and feasibility study included qualitative assessments with patients and clinicians that highlight the need to enhance the flow of real time data shared with the care team and the need to integrate within the care team work flow including real time data sharing of the patient's app data within the EMR<sup>16</sup>. It also highlighted the need for care team education on measurement-based care, shared-decision making, and collaborative care and on how to utilize the Pathway App to improve these processes. Building on these results we created the *Pathway Platform* which includes a newer iteration of the Pathway App along with real time patient level data shared with the EMR integration in real-time and educational program both care team and patient facing.

We aim to implement a digitally enabled care pathway referred to as the *Pathway Platform* and assess its impact on measurement-based care and other evidence-based processes. The primary objective is to determine whether PHQ-9 utilization, a measurement- based practice, is greater after is the Pathway Platform implemented.

#### 3. STUDY DESIGN

We will use a pre- post- study design to assess the impact of implementing the Pathway Platform in the primary care setting. Clinic performance and select patient outcomes will be compared before and after implementation. Additional patient outcomes will be assessed after implementation among patients using the Pathway Platform (**Figure 1**).

This study will be performed within primary care clinics in Advocate's Health Care System. Advocate is the largest healthcare provider in the state of Illinois with 12 hospitals, 20 health centers, and 250+ care sites. It is one of the largest Accountable Care Organizations in the United States caring for over 2 million patients annually. General practitioners provide diagnoses, treatment, and clinical care for adults ages 18 and over with chronic diseases, which often includes MDD.

#### 3.1 Performance among participating clinics post-implementation

The Pathway Platform will be implemented in up to 20 primary care sites within the Advocate Aurora Health system and enroll a total of 200 patients for six-month duration. The visit where the patient has been onboarded to the Pathway Platform will be the enrollment visit (Figure 1). During the post- implementation period, data on patient outcomes will be collected through the Pathway Platform. At the end of the study an electronic and manual chart review for patients using the Pathway Platform will be conducted among participating clinics and performance related to measurement-based care, shared decision making and collaborative care, where applicable, will be assessed over the post-implementation period.

# 3.2 Retrospective Assessment: pre-implementation performance at the clinic level (before Pathway Platform implementation)

To assess Advocate's primary care sites performance pre-implementation, an electronic and manual chart review will be conducted from the same Advocate primary care clinics participating in the implementation study. Patients with a clinic visit at least 6 months prior to implementation (index visit) of the Pathway Platform and meeting the inclusion criteria for enrollment in the study, will be included in this analysis (figure 1). Patient history will be evaluated for three months prior to index visit to confirm eligibility. The goal is to capture patients with a new start, dose adjustment or switch of an antidepressant medication 6 months prior to the implementation index date (three-month inclusion window for patient identification). Six months of patient history will be "retrospectively" collected for this baseline patient cohort to assess the primary outcome, defined as PHQ-9 utilization, and other secondary outcomes outlined in the protocol. This analysis will serve as the comparison control for the primary and secondary outcomes to compare performance at the same clinics pre and post-implementation of the Pathway Platform. Depending on the number of eligible patients identified per site (20 per site), group level matching for age and sex may be conducted. The primary endpoint will be the proportion of patients with at least 2 PHQ-9 scores.



\* Primary and secondary outcomes will be evaluated at 6 months, data collected beyond 6 months will be used for exploratory analysis

#### 4. SELECTION AND ENROLLMENT OF PARTICIPANTS

Patients will be recruited from up to 20 primary care clinics within Advocate Aurora Health that have agreed to implement the Pathway Platform. We aim to identify clinics that are representative of different geographic locations, patient populations, and care models for depression management, including behavioral health integration models. We will balance clinic diversity with feasibility to conduct this study. For example, we will only include clinics that have integrated Epic within their workflow so that the care team can easily access data collected from the patient in the Pathway Platform. We will also focus on clinics that have a large volume of patients diagnosed with depression as well as clinics that have care team members that are interested and engaged in depression care.

All care team members who care for patients with depression will be invited to participate in this implementation study and will have access to an online educational resource center. Patients fulfilling the following criteria will be eligible to download and use the Pathway Platform:

#### 4.1 Inclusion

1. Adult aged 18 and above

- 2. Diagnosis with major depressive disorder or reference to "clinical depression" in patient charts. See **Appendix 1** for ICD codes for major depressive disorders
- 3. Recently prescribed monotherapy antidepressant medication (defined as new start, medication switch, or dose change in the past 3 months (**Appendix 2**).
- 4. Patients with inadequate response or tolerability concerns determined based on A PHQ-2 score of 3 or greater, or a PHQ-2 <3 with a PHQ-9 score of 5 or greater recorded in medical records in the past 6 weeks or during screening,
- 5. Able and willing to provide informed consent
- 6. Able to use the Pathway Platform based on clinician's judgment, e.g. owns an iPhone version 5 or later or smartphones with Android operating systems, have an active data plan or regular WiFi access.

#### 4.2 Exclusion

- 1. Missing PHQ-2/PHQ-9 score in the past 6 weeks and/or unable to perform PHQ-2/PHQ-9 at index visit
- 2. Diagnosis with bipolar depression, schizophrenia, and/or schizoaffective disorder, (Appendix 1).
- 3. Patient no longer under primary care for depression and has transitioned to a psychiatric care team (i.e., Psychiatrist, Advance Practice Psychiatric Nurse, Psychiatric Nurse Practitioner, Psychiatric Physician Assistant).
- 4. Lack of functional English literacy (indicated by primary language in EMR).

#### 4.3 Study Enrollment Procedures

This is a real-world implementation study with minimal interaction between the study team and patients. To address recent virtual visits in primary care due to COVID-19 and for the safety of the study team, study methods were developed to adapt virtual patient recruitment and e-consent during existing virtual visit processes. An in person consenting process is also available for in person clinic visits, when safe and appropriate, and will be supported by a study team member present at recruiting clinics.

Study team will review clinic schedules routinely for visits scheduled the next day and will flag potentially eligible patients and will discuss the list with the health care team. These patients will be introduced to the study opportunity by care team members during routine clinic visits.

- Consenting in person: If the patient is interested, they will be roomed with a study team member who will confirm study eligibility and provide written informed consent. If the patient is eligible and provides consent, the study team will share a secure message with a link for the Pathway App with the patient and the patient will be able to activate the Pathway App and start entering data. The secure message will be shared with the patient via AAH's secure patient portal. Or through an email for patients who have not activated their portal. The invitation message in the email will include an individualized link to download the App with a unique code specific to that patient to ensure security.
- e-Consenting virtually: If the patient is interested, the care team member will inform the research team, who will confirm eligibility and send a secure invitation to the patient (AAH patient portal or email with unique link and code). The invitation message includes a link to start the e-consenting process and that includes study contact information to allow patients to reach out to the study team with any questions during e-consenting or during the study. The link in the message will direct the patient to start the e-consenting process. The patient will not be able to download the app until they have completed the e-consenting process. Patient e-consent will be obtained in REDCap using a finger or stylus-directed signature on the mobile phone, with data including attestation of individual identity and time and date of signing. Upon completion, participants will be able to download a pdf copy of the signed e-consent form. The patient will then be invited to download the Pathway App via another secure message with a link including details for the patient to activate the mobile app and start entering data.

#### 4.4 Pathway Platform

The Pathway Platform consists of three components:

#### 4.4.1 Pathway App

Pathway is a mobile application designed to gather health information related to the management of depression to enhance patient clinical engagement and guide patient care. The patient facing interface includes a digital assistant that allows patients to interact with the Pathway Platform in a chat-based conversational text interface. The information collected from the patient is intended to assist the care team in managing the patient's depression through enhancing measurement-based care and shared-decision making - enhancing patient-provider engagement and ultimately patient outcomes. The study will deploy the most recent iteration of the Pathway Platform. Earlier iterations were piloted in four primary care clinics. <sup>16</sup> Feedback from this pilot was used to enhance Pathway Platform functionality. The current iteration of the Pathway Platform, which is the version that will be used in the implementation study described in this protocol, prompts patients to complete four scales to assess depression status biweekly (Patient Health Questionnaire [PHQ-9] and Perceived Deficits Questionnaire-Depression [PDQ-D5]), quality of life (World Health Organization- Five Well Being Index [WHO-5]), and cognition (Digit Symbol Substitution Test [DSST]). 7,17,18,19 The Pathway Platform also includes a daily evening check-in with the patient to collect information on medication adherence and side effects. Patients reporting side effects related to sleep are prompted to complete the PROMIS Sleep Disturbance 6a and patients reporting side effects related to sexual dysfunction are prompted to complete the Arizona Sexual Experience Scale (ASEX).<sup>20,21</sup> An optional functionality of the Pathway Platform is to set and track goals using the Goal Attainment approach adapted for depression during clinic visits with a healthcare provider.<sup>22</sup> In addition, the Pathway Platform includes patient facing education for the patient on how to use the Pathway Platform to collect data as well as how to prepare for a visit with health care providers, set and assess progress towards goals and self-management. For purposes of evaluating this implementation study three additional scales assessing patient-provider engagement and functional improvement will be deployed through the Pathway Platform at baseline and subsequently every 6 months until the end of the study (Patient Activation Measure -13[PAM-13], CollaboRATE, and Work and Social Adjustment Scale [WSAS]). 23,24,25

#### 4.4.2 Electronic Medical Record integration

Data collected in the Pathway Platform is electronically transmitted and stored in the patient's EMR. This data is accessible to the care team and provides a longitudinal summary that may assist in decision making and depression management. Providers can view this data either before or during the patient visit and use it to discuss future depression management.

#### 4.4.3 Educational Scaffolding

An online Educational training program was developed using evidence-based medicine building

on measurement-based care and shared-decision making concepts as they relate to depression management. Educational material describes how the Pathway Platform can help care team members in clinical processes related to these process improvement measures. In clinics using a collaborative care model additional education material specific to this care model is provided. Educational material housed in an online resource center which includes reading material, presentations, and videos. Additionally, up to three audit and feedback sessions will be conducted for each participating clinic. The objectives of audit and feedback sessions are to benchmark performance measures, including shared decision making, reflect on current clinical practice and improvement strategies, and setting team-based action plans. Care team members who manage depression must complete specific training before they are able to enroll patients and begin using the Pathway Platform.

A training manual was also developed for patients. The manual describes the Pathway Platform functionality, as well as, how to use and interpret the data collected.

#### 3.3 Study Duration

Patients will be enrolled in the study for a minimum duration of 6 months with the option to continue using the app at that time to a common study end date of January 7, 2023 (access to inapp final study evaluations will end January 21, 2023). Data from the Pathway Platform will be collected prospectively for the duration of the patient's participation. Process measures will be collected retrospectively from the EMR and through manual chart review after 6 months of enrollment and at the end of the study(post-implementation) and over a 6-month period prior to implementation (pre-implementation).

#### 5. STUDY PROCEDURES

#### 5.1 Schedule of events

| Table 1: Schedule of evaluations | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Pre-<br>electronic<br>and<br>manual<br>chart<br>reviews | Complete<br>education<br>by care<br>team | Screening | Baseline<br>assessment | | Assessment | Final assessment | |
| Study Day/Week: | | Day -1 | Day 0 | Day 1 | Day 168 | 8 - 172^ | Stud | ly end |
| Visit Windows (Days): | | | | | | | | |
| Source | | | EMR/<br>patient<br>scheduling | Pathway<br>Platform | Pathway<br>Platform | EMR and<br>Manual<br>Review | Pathway<br>Platform | EMR and<br>Manual<br>Review |
| Patient electronic screening | | | X | | | | | |
| Informed consent | | | X | | | | | |
| Onboarding | | | X | | | | | |
| Demographic characteristics | X | | | | | | | |
| Number of PHQ-9 scores documented | X | | | | X | X | X | X |
| Treatment adjustments | X | | | | X | X | X | X |
| Shared decision making (OPTION-12 and CollaboRATE) | X | | | | X | X | X | X |
| Referral to behavioral health | X | | | | | X | | X |
| PHQ-9 scores | X | | | | X | | X | |
| Emergency room visits | X | | | | | X | | X |
| Emergency room visits due to mental illness | X | | | | | X | | X |
| Hospital admissions | X | | | | | X | | X |
| Follow up after emergency room and | X | | | | | X | | X |
| hospital visits | Λ | | | | | A | | Λ |
| Hospital admissions due to mental illness | X | | | | | X | | X |
| Healthcare resource utilization | | | | | | | | |
| Outpatient visits including phone calls | X | | | | | v | | X |
| Outpatient visits including phone calls | X | | | | | X<br>X | | X |
| due to mental illness | Λ | | | | | Λ | | Λ |
| | 37 | | | | v | | V | |
| Remission and response (using PHQ-9 data) | X | | | | X | | X | |
| PAM 13 *** | | | | X | X | | X | |
| CollaboRATE**, *** | | | | X | X | | X | |
| WSAS *** | | | | X | X | | X | |
| PHQ-9 | | | | X | X | X | X | X |
| WHO-5 | | | | X | X | | X | |
| PDQ-D5 | | | | X | X | | X | |
| Medication adherence | | | | X | X | | X | |
| Side effects | | | | X | X | | X | |
| PSD-6 (only if reporting side effects of sleep problems) | | | | X | X | | X | |
| ASEX (only if reporting side effects of sexual problems) | | | | X | X | | X | |
| Goal Setting | | | | X | | | | |
| Goal Attainment | | | | 11 | X | | X | |
| App analytics | | | | X | X | | X | |
| Report analytics | | | | X | X | | X | |
| Educational material analytics | | | | X | X | | X | |
| In depth interviews (Patients and | | | | Λ | Λ | | X | |
| Clinicians) | | | | | | | | |
| Adverse Events* | X | | X | X | X | | X | X |
| Serious Adverse Events | X | | X | X | X | | X | X |
| ^Day 168 reflects and of initial 24 week | | المالم الماليات الماليات | final act of | | | la for complation | (DIIO O III | 110.51 |

<sup>^</sup>Day 168 reflects end of initial 24 week study period in which the final set of care questionnaires are available for completion (PHQ-9, WHO-5 and PDQ-D5), these expire within 3 days. Day 172; The off-boarding process is available, including the research questions (PAM-13, WSAS,

CollaboRATE), these expire after 30 days.

\*If during the conduct of the study, a health care professional or patient spontaneously reports an Adverse Event or a serious adverse event to a Takeda product; such information should be reported to the sponsor. As such reports are spontaneously notified, causality of any AEs should be assumed unless there is evidence to the contrary; \*\*CollaboRATE will also be asked within the App at Day 84 with a 30 day window for completion during patient enrollment. \*\*\*PAM 13, CollaboRATE and WSAS; the App will trigger response to these questionnaires every 6 months until study end (note; if patient completed these questionnaires within 4 weeks of study end point, they will not be re-deployed for completion at end of study).

#### 5.2 Description of study evaluations

- 1. EMR data pulls and manual chart reviews: EMR data and manual chart review data will be collected from two cohorts of patients: (1) patients attending clinics after implementation (post- implementation cohort) and (2) patients attending clinics before implementation (pre-implementation). For the pre-implementation cohort, data will be collected over a sixmonth period. For the post-implementation cohort, data will be collected from the time of study implementation until the end of the study.
- 2. Pathway Platform data and analytics: Data on patient outcomes and Pathway Platform usage will be collected throughout the study starting at day 1 and ending on the final day of the patient's participation (i.e. 6 months, common study end date or patient withdrawl). Similarly, data on report usage by care team will be collected throughout the study.
- 3. Educational resource center analytics: The number of times material in the resource center is viewed will be recorded between day 1 and the end of the study.

#### 6. SAFETY ASSESSMENTS

#### 6.1 Adverse Events Related to the Pathway Platform

No adverse events (AEs) are expected in this minimal risk study related to the Pathway Platform; however, all serious adverse events (SAEs) that are spontaneously reported during the study period will be collected.

A SAE is defined as an adverse event, reported during the implementation study of the Pathway Platform, in the view of either the investigator or sponsor, results in any of the following outcomes:

- a. Death
- b. Life-threatening adverse event
- c. Inpatient hospitalization or prolongation of existing hospitalization (for > 24 hours)
- d. Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- e. Congenital anomaly/birth defect.

f. Important medical events that may not result in death, be life-threatening or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

The following information will be collected for any SAE that is reported:

- Event details
- Start and stop date
- Frequency
- Intensity
- Investigator's opinion of the causal relationship to study procedure(s), including the details of the suspected procedure
- Outcome of event
- Severity

Causality to study procedures will be determined for all SAEs and deemed "related" or "not related" to the intervention. Severity will be assessed as mild (event is transient and easily tolerated by the subject), moderate (event causes the subject discomfort and interrupts the subjects' usual activities), or severe (event causes considerable interference with the subject's usual activities). The start date of the SAE is the date that the first signs or symptoms were noted. The stop date is the date on which the subject recovered, the event resolved, or the subject died.

All SAEs, along with the information bulleted above, will be compiled and included in the final study report. SAEs will be reported to Takeda within 24 hours of becoming aware of the event.

#### 6.2 Change in Participant Suicidal Ideation

Patients using the Pathway Platform will answer biweekly PHQ-9 surveys, during which Item 9 asks about the frequency of suicidal ideation. It is possible that a patient will report a change in suicidal ideation in the course of responding to this question. In the event that a patient responds affirmatively to this question, the patient will receive a pop-up notification that s/he should contact his/her health care provider or emergency services immediately. This instruction is what is given in routine clinical practice. The

data from the Pathway Platform is not monitored in real time by care teams. Patients will be informed via consent that the information provided to the Pathway Platform is not directly or continuously monitored. As an additional item of note, data from the Pathway Platform may be delayed and/or not received by the EMR if device is unable to transmit data.

This information will also be included in the patient consent and will be explained to the patient by the Care Team during the consent process.

#### 7. INTERVENTION DISCONTINUATION

Patients are not required to use the Pathway Platform and can choose to discontinue at any time. Adherence to use will be tracked and reported for analytical purposes.

#### 8. STATISTICAL CONSIDERATIONS

#### 8.1 General Design and Hypothesis

The following hypotheses will be examined:

Primary hypothesis: PHQ-9 utilization will be greater after implementation compared to before implementation of the Pathway Platform.

Secondary hypothesis: Provider processes and patient depression related outcomes will have greater improvements in patient outcomes after implementation of the App compared to previous practice patterns.

#### 8.2 Sample size and randomization

The primary outcome for this study is PHQ-9 utilization. Assuming 75% PHQ-9 utilization prior to implementation of the Pathway Platform and 90% PHQ-9 utilization after implementation of the Pathway Platform, we will need 100 patients per group, for a total of 200 patients, assuming 80% power and a 2-sided alpha of 0.05 using Pearson chi square test for two independent proportions. To allow for subgroup analyses the sample will include 200 patients per group, for a total of 400 patients; 200 patients will comprise the "post-implementation" cohort and 200 will comprise the "pre-implementation" cohort. **Table 2** presents additional sample size calculations based on different assumptions of PHQ-9 utilization.

**Table 2**: Sample size calculations based on different assumptions of PHQ-9 utilization, alpha = 0.05, Power = 80%.

| PHQ-9 | utilization | pre- | PHQ-9 in | Pathway | post- | N patients per group |
|---|---|---|---|---|---|---|
| implement | tation | | implementa | tion | | |
| 75% | | | 80% | | | 1,094 per group |
| 75% | | | 90% | | | 100 per group |
| 75% | | | 95% | | | 49 per group |
| 50% | | | 65% | | | 170 per group |
| 50% | | | 80% | | • | 30 per group |
| 50% | | • | 90% | | • | 20 er group |

#### 8.3 Outcomes

#### 8.3.1 Primary outcome

The primary process outcome is PHQ-9 utilization over a six-month period. For purposes of this study, PHQ-9 utilization will be defined as documentation of at least 2 PHQ-9 scores in the EMR over the initial 6-month study period. The proportion of patients who meet this definition will be compared between patients attending clinics pre- and post- implementation of the Pathway Platform. Additional analyses exploring the number of PHQ-9s over the study period will also be conducted.

#### 8.3.2 Secondary outcome

*Process outcomes*: The following secondary process outcomes will be compared between patients attending clinics pre- and post- implementation of the Pathway Platform.

- Measurement- based care: The proportion of patients reflecting measurement-based care
  informed MDD treatment adjustments in their charts, defined as at least one dose change,
  medication switch, or add on medication during the study period. The frequency and types
  of treatment adjustments will also be explored.
- Shared- decision making: The proportion of patients reflecting shared-decision making, using the OPTION12 Tool framework.<sup>26</sup> The tool will be modified by adding a thirteenth domain inquiring about goal setting (Asking the patient or caregiver about goals of treatment). The frequency and domains of shared-decision making will also be explored in a manual chart review and a variable added to assess if the clinician documented asking the patient about their goals of treatment.
- Referrals to behavioral health: The proportion of patients with at least one referral will be compared. The frequency and types of referrals will also be explored.
- Follow-up after hospitalization for mental illness: The proportion of hospitalized adults who receive follow-up within 7 days of discharge and within 30 days of discharge.
- Follow-up after emergency department visit for mental illness: The proportion of adults

- who receive follow-up within 7 days of discharge and within 30 days of ED visit.
- Healthcare resource utilization: Number and costs associated with hospital admission, length of stay, emergency room admissions, and encounters with outpatient clinics. Costs will be calculated using USA national average costs for inpatient and outpatient visits or using an average Advocate Health Care system cost.

Patient clinical outcomes: The following outcomes will be compared between patients attending clinics pre- and post- implementation of the Pathway Platform, keeping in mind that the number of patients with these measures in the pre- implementation patient group will be limited:

- MDD remission: The proportion of patients with PHQ-9 <= 5 at the end of the study period. The last measurement available during the study period will be used to calculate remission.
- MDD response: The proportion of patients with a 50% or greater reduction in PHQ-9 scores. The first and last scores available during the study period will be used to calculate response.
- Diagnosis progress notes stating change from mild, moderate, or sever, to in remission or partial remission will be assessed descriptively.

*Patient reported outcomes*: The difference in scores between baseline, and 6-month follow up will be compared among patients using the Pathway Platform who completed the following measures:

- PAM-13
- CollaboRATE (this questionnaire is also included as a 3-month post-enrollment assessment and will be analyzed across all available time points)
- WSAS

#### 8.3.3 Exploratory outcomes

Patient clinical and reported outcomes:

- The following patient reported outcomes will be collected in the Pathway Platform throughout the study. The difference in scores between the baseline measure, 6-months, and end of the studywill be compared. This will be restricted to patients who completed these scales at these two-time points. To be inclusive of all patients, additional analyses will be conducted to compare first and last scores available:
  - o PHQ-9
  - o WHO-5
  - o PDQ-D5

- The following patient reported outcomes will be collected in the Pathway Platform and described at 6-months and end of the study:
  - Antidepressant Medication adherence
  - o Antidepressant Medication dose adjustment and switches
  - Side effects
  - Depression remission
  - Depression response
  - o Goal attainment
  - Patient reported outcomes (PAM-13, CollaboRATE and WSAS) will also be explored at 6 months and end of the study.

Pathway Platform and report utilization: Pathway Platform analytics will be explored to understand patient adherence to the platform which includes frequency of logging into the Pathway Platform and frequency of completing each of the Pathway Platform functionalities. Care-team utilization of Pathway Platform reports will also be explored, including describing type of care team members who viewed the Pathway Platform reports as well as frequency of viewing the reports.

*Education utilization:* Frequency of viewing material in the resource education center will be described by patient and by care-team members. Commonly viewed educational material will be highlighted.

Subgroup analysis: primary, secondary, and exploratory outcomes will be compared across a number of patient demographic and clinical characteristics, including PHQ-9 severity at baseline, comorbidities (see appendix 3 for comorbid conditions and ICD codes), app utilization by patients, and EMR report utilization by providers. Additional subgroup analysis will be conducted by type of care model at the site level (e.g. collaborative care vs. non collaborative care sites).

#### 8.3.4 Patient and provider in-depth interviews

In-depth interviews will be conducted at the end of the study period with approximately 20 patients and 15 care team members who have used the Pathway Platform. Interviews will involve discussing reactions and feedback on the Pathway Platform, education material, care team interface, and overall implementation of the Pathway Platform. These semi-instructed in-depth interviews will allow patients to reflect on the process and identify higher level causes behind any difficulties or challenges, explore any suggested changes and to gather general feedback regarding the participant's experience during the study. Findings from this sub-study will complement the main study analysis and explore the use of the Pathway Platform App and what this could mean for ongoing development of the Pathway Platform.

#### 8.3.5 System level performance

Performance and patient outcomes evaluated in this study will be evaluated at the system level covering all primary care clinics. Data will be collected retrospectively on patients attending any primary care clinic during the study period. This data will be used to understand performance at the system level.

#### 8.4 Data analysis

**For primary and secondary hypothesis testing**, process measures, patient clinical outcomes, and health care resource utilization will be compared pre- and post- implementation of the Pathway Platform.

Additional patient reported outcomes will be compared among patients using the Pathway Platform only at baseline and end of study. For pre-implementation, outcomes will be assessed among patients who visited one of the study clinics at least once over the pre-implementation study period and were eligible to use the Pathway Platform, if it had been available. For the post-implementation period, the Pathway Platform will be the data source for paired t-test analysis, assessing change in continuous variables including PHQ-9 scores. Categorical outcomes will be presented as proportions and compared using Pearson Chi2 test. Continuous outcomes will be assessed for normality and presented as means and standard deviations (SD) or medians and interquartile ranges (IQR); continuous outcomes will be compared using Student's t test for independent groups. Two-tailed tests using a significance threshold of p < 0.05 will be used for all tests.

**Exploratory outcomes**: will be described among patients attending the pathway platform clinics only and will be compared between baseline, 6-month and extended follow up. Change in these outcomes overtime, including utilization analytics will also be explored. Categorical outcomes will be presented as proportions and compared using McNemars' test. Continuous outcomes will be assessed for normality and presented as means and standard deviations (SD) or medians and interquartile ranges (IQR); continuous outcomes will be compared using Student's Paired t test for single group comparison. Two-tailed tests using a significance threshold of p < 0.05 will be used for all tests. Goal attainment will be summarized by proportion of patients who achieve their identified goals based on the set time bound duration of the goal (i.e., GAS Score  $\geq$ 50).  $^{29,30}$  The goal attainment scale adapted for depression yields a norm-based score (standardized to a mean of 50, SD of 10) at baseline and at the end of the time bound goal; the change from score from baseline will also be summarized.

**System level performance**: Process outcomes will be evaluated at the system level (all primary

care clinics) among patients fulfilling eligibility criteria, if the app were available. Descriptive analysis will be utilized to describe process outcomes across all clinics.

In depth interviews: Interpretative Phenomenological Analysis will be used to analyze the qualitative data. To increase the rigor and validity of the analysis, and as a form of triangulation, the analysis will be conducted by 3 members of the research team (the lead qualitative researcher and 2 others). Analysis will involve 2 stages: (1) Data management, which will include, familiarization with the data, reading notes, and/or listening to the audio dialogue in order to extract main themes and ideas and thematic framework development, identifying the key issues and concepts present in the data and creating themes both inductively, based on the data, and deductively, based on the research questions, (2) Interpretation stage, which will include focused defining the main concepts and mapping the ways in which different parts of the data are related to each other.

#### 4. 9.4 PARTICIPANT RIGHTS AND CONFIDENTIALITY

#### 4.1 9.4.1 Institutional Review Board (IRB) Review

This protocol, the informed consent document, and any subsequent modifications will be reviewed and approved by the Advocate's IRB, who is responsible for oversight of the study.

#### 4.2 **9.4.2** Informed Consent Forms

A signed consent form will be obtained from each participant by the Advocate Research Team. The consent form will describe the purpose of the study, the procedures to be followed, and the risks and benefits of participation. A copy will be given to each participant and will be documented in the participant's record.

#### 4.3 **9.4.3** Participant Confidentiality

Data will be extracted from an EMR data pull as well as chart reviews and shared only with the clinic and research staff that are needed to identify eligible patients for the study in a password-protected MS Excel sheet. For clinic staff, shared patient information will be limited to only the patients seen at that clinic location. All paper copies of study data collection forms will be stored in a secure location at Advocate Research Institute to maintain subject confidentiality.

A subject ID will be assigned to each study participant; this will serve as a unique subject identifier for the study and Pathway Platform data. Data management for Pathway Platform data will have security processes in place that are service organizational control

or SOC2 compliant. This comprises data storage and transmission between the Pathway Platform, servers, and EMR system. Data collected for the study will be maintained and monitored while the study is active and the identifying link will be destroyed upon study close.

#### 4.4 **9.4.4Study Discontinuation**

The study may be discontinued at any time to ensure that research patients are protected.

## 5. 10. TAKEDA MARKETED PRODUCT ADVERSE EVENT REPORTING REQUIREMENTS

An AE is any untoward medical occurrence in a subject administered a Takeda medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a Takeda medicinal product, whether the event is considered causally related to the use of the Takeda product.

#### 10.1 Special Situation Reports and Product Quality Issues

A special situation report (SSR) includes any of the following events:

- Pregnancy: Any case in which a pregnant patient is exposed to a Takeda product or in which a female patient or female partner of a male patient becomes pregnant following treatment with Takeda product. Exposure is considered either through maternal exposure or via semen following paternal exposure.
- Breastfeeding: Infant exposure from breast milk.
- Overdose: All information of any accidental or intentional overdose.
- Drug abuse, misuse or medication error: All information on medicinal product abuse, misuse or medication error (potential or actual).
- Suspected transmission of an infectious agent: All information on a suspected (in the sense of confirmed or potential) transmission of an infectious agent by a medicinal product.
- Lack of efficacy of Takeda product.
- Occupational exposure.
- Use outside the terms of the marketing authorization, also known as "off-label".
- Use of falsified medicinal product.

A product quality issue refers to defects related to the safety, identity, strength, quality, or purity of the product or with the physical characteristics, packaging, labeling, or design of the product.

#### 10.2 Procedures

Collection and Reporting of Spontaneous AEs, SSRs, and Product Quality Issues Related to a Takeda Product: If during the conduct of the study, a health care professional or patient spontaneously reports an AE, SSR, or product quality issue where the event/issue pertains to a Takeda product (or unbranded generic); such information should be reported to the sponsor. As such reports are spontaneously notified, causality of any AEs should be assumed unless there is evidence to the contrary.

AEs, SSRs or products complaints relating to any Takeda products received spontaneously must be reported via email or by telephone within 24 hours of awareness and no later than by the next working day. The preferred method for reporting is via email. If a report is received via telephone it should be backed up with an email. Advocate may submit Reportable Information to Takeda at <a href="mailto:medicalinformation@tpna.com">medicalinformation@tpna.com</a>. Alternatively, Advocate may submit Reportable Information to Takeda's Call Center by calling 1-877-Takeda7.

#### 6. 11. PUBLICATION OF RESEARCH FINDINGS

Publication of the results of this study will be governed by the policies and procedures developed by the Steering Committee, which will include representatives from Advocate Health Care and the Takeda/Lundbeck Alliance. Any presentation, abstract, or manuscript related to the data resulting from this study will be made available for review by Advocate Health Care and the Takeda/Lundbeck Alliance prior to submission.

#### 7. REFERENCES

- 1. van Os J, Delespaul P, Barge D, Bakker RP. Testing an mHealth momentary assessment Routine Outcome Monitoring application: a focus on restoration of daily life positive mood states. *PloS one*. 2014;9(12):e115254
- 2. Robotham D, Satkunanathan S, Doughty L, Wykes T. Do We Still Have a Digital Divide in Mental Health? A Five-Year Survey Follow-up. *J Med Internet Res.* 2016;18(11):e309.
- 3. Trivedi MH, Jha MK, Kahalnik F, Pipes R, Levinson S, Lawson T, Rush AJ, Trombello JM, Grannemann B, Tovian C, Kinney R, Clark EW and Greer TL. VitalSign. A Primary Care First (PCP-First) Model for Universal Screening and Measurement-Based Care for Depression. *Pharmaceuticals (Basel, Switzerland)*, *12*(2), 71. doi:10.3390/ph12020071
- 4. Rathbone, A. L., & Prescott, J. (2017). The Use of Mobile Apps and SMS Messaging as Physical and Mental Health Interventions: Systematic Review. *Journal of medical Internet research*, *19*(8), e295. doi:10.2196/jmir.7740

- 5. Silverman JJ, Galanter M, Jackson-Triche M, Jacobs DG, Lomax JW, Riba MB, Tong LD, Watkins KE, Fochtmann LJ, Rhoads RS, Yager J and Association AP. The American Psychiatric Association Practice Guidelines for the Psychiatric Evaluation of Adults. *Am J Psychiatry*. 2015;172:798-802.
- 6. Torous J, Staples P, Shanahan M, Lin C, Peck P, Keshavan M and Onnela JP. Utilizing a Personal Smartphone Custom App to Assess the Patient Health Questionnaire-9 (PHQ-9) Depressive Symptoms in Patients With Major Depressive Disorder. *JMIR Ment Health*. 2015;2:e8.
- 7. Kroenke K, Spitzer RL and Williams JB. The PHQ-9: validity of a brief depression severity measure. *J Gen Intern Med*. 2001;16:606-13.
- 8. Loh A, Simon D, Wills CE, Kriston L, Niebling W and Härter M. The effects of a shared decision-making intervention in primary care of depression: a cluster-randomized controlled trial. *Patient Educ Couns.* 2007;67:324-32.
- 9. Hopwood M. The Shared Decision-Making Process in the Pharmacological Management of Depression. *Patient*. 2019.
- 10. Von Korff M, Gruman J, Schaefer J, Curry SJ and Wagner EH. Collaborative management of chronic illness. *Ann Intern Med.* 1997;127:1097-102.
- 11. Katon WRobinson PVonKorff MLin EBush TLudman ESimon GWalker GA multifaceted intervention to improve treatment of depression in primary care. *Arch Gen Psychiatry*. 1996;53924-932
- 12. Organization WH. Depression: A Global Public Health Concern. 2012. Accessed February 28, 2019.
- 13. McIntyre RS, Cha DS, Soczynska JK, et al. Cognitive deficits and functional outcomes in major depressive disorder: determinants, substrates, and treatment interventions. *Depress Anxiety*. 2013;30(6):515-527.
- 14. Greenberg PE, Fournier AA, Sisitsky T, Pike CT, Kessler RC. The economic burden of adults with major depressive disorder in the United States (2005 and 2010). *The Journal of clinical psychiatry*. 2015;76(2):155-162.
- 15. Kessler RC, Merikangas KR, Wang PS. The prevalence and correlates of workplace depression in the national comorbidity survey replication. *Journal of occupational and environmental medicine*. 2008;50(4):381-390.
- 16. Maggie McCue, Christopher Blair, Ben Fehnert, Francesca Cormack, Sara Sarkey, Anna Eramo, Ellen Rhodes, Christopher Kabir, Rasha Khatib, David Kemp. A Collaborative Study to Assess Digitally Enabled Engagement in Major Depressive Disorder Within a Large Health System. APA, San Francisco, CA; May 2019.

- 17. Lam R, Saragoussi D, Danchenko N, Lamy F, Rive B, Brevig T. Psychometric validation of Perceived Deficits Questionnaire Depression (PDQ-D) in patients with major depressive disorder. Value in Health 2013;16(7):A330. ISPOR 16th Annual European Congress, Poster QL4.
- 18. Wellbeing Measures in Primary Health Care/The Depcare Project. WHO Regional Office for Europe. 12-13 February 1998. Publication No. EUR/ICP/QCPH 05 01 03.
- 19. Wechsler D. Adult Intelligence Scale. 3rd ed. San Antonio, TX: Psychological Corporation: 1997.
- 20. Buysse DJ, Yu L, Moul DE, et al. Development and Validation of Patient-Reported Outcome Measures for Sleep Disturbance and Sleep-Related Impairments. *Sleep*. 2010;33(6): 781–792
- 21. McGahuey CA, Gelenberg AJ, Laukes CA et al. The Arizona Sexual Experience Scale (ASEX): reliability and validity. Journal of Sex & Amp; Marital Therapy. 2000;26:25-40.
- 22. McCue M, Parikh SV, Mucha L, Sarkey S, Cao C, Eramo A, Opler M, Webber-Lind B, François C.Adapting the Goal Attainment Approach for Major Depressive Disorder. Neurol Ther. 2019 Aug 21. doi: 10.1007/s40120-019-00151-w.
- 23. Hibbard, J.H., Mahoney E.R., Stockard J., and Tusler M. Development and Testing of a Short Form of the Patient Activation Measure. Health Services Research 40:6, Part I (December 2005).
- 24. Forcino RC, Barr PJ, O'Malley AJ, et al. Using CollaboRATE, a brief patient-reported measure of shared decision making: Results from three clinical settings in the United States. Health Expect. 2018;21(1):82–89. doi:10.1111/hex.12588
- 25. Mundt JC, Marks IM, Shear MK, Greist JM. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. British Journal of Psychiatry. 2002;180(5):461-464. doi:10.1192/bjp.180.5.461
- 26. Elwyn G, Edwards A, Wensing M, *et al.* Shared decision making: developing the OPTION scale for measuring patient involvement. BMJ Quality & Safety 2003;12:93-99.
- 27. Elwyn G, Edwards A, Kinnersley P, Grol R. Shared decision making and the concept of equipoise: the competences of involving patients in healthcare choices. Br J Gen Pract. 2000 Nov;50(460):892-9.
- 28. Elwyn,G, Edwards, A, Wensing, M, Grol, R. Shared decision making measurement using the OPTION instrument.

- 29. Kiresuk TJ, Sherman RE. Goal attainment scaling: A general method for evaluating comprehensive community mental health programs. Community Ment Health J 1968;4(6):443-53
- 30. McCue M, Parikh SV, Mucha L, et al. Personalized Goal Attainment After a Switch to Vortioxetine in Adults With Major Depressive Disorder (MDD): Results of a Phase 4, Open-Label Clinical Trial. Poster presented at: Psych Congress; 2018 Oct 25 Oct 28; Orlando, FL.

| Appendix 1: Se | Appendix 1: Selection criteria ICD codes | |
|---|---|---|
| Code Type | Code | Description |
| ICD-9-CM DX | 296.26 | Major depressive disorder, single episode in full remission |
| ICD-9-CM DX | 296.25 | Major depressive disorder, single episode, in partial or unspecified remission |
| ICD-9-CM DX | 296.21 | Major depressive disorder, single episode, mild |
| ICD-9-CM DX | 296.22 | Major depressive disorder, single episode, moderate |
| ICD-9-CM DX | 296.24 | Major depressive disorder, single episode, severe, specified as with psychotic behavior |
| ICD-9-CM DX | 296.23 | Major depressive disorder, single episode, severe, without mention of psychotic behavior |
| ICD-9-CM DX | 296.20 | Major depressive disorder, single episode, unspecified |
| ICD-9-CM DX | 296.36 | Major depressive disorder, recurrent episode, in full remission |
| ICD-9-CM DX | 296.35 | Major depressive disorder, recurrent episode, in partial or unspecified remission |
| ICD-9-CM DX | 296.31 | Major depressive disorder, recurrent episode, mild |
| ICD-9-CM DX | 296.32 | Major depressive disorder, recurrent episode, moderate |
| ICD-9-CM DX | 296.34 | Major depressive disorder, recurrent episode, severe, specified as with psychotic behavior |
| ICD-9-CM DX | 296.33 | Major depressive disorder, recurrent episode, severe, without mention of psychotic behavior |
| ICD-9-CM DX | 296.30 | Major depressive disorder, recurrent episode, unspecified |
| ICD-9-CM DX | 296.x | Manic depression/bipolar disorder (Episodic Mood Disorder) |
| ICD-9-CM DX | 295.9x | Schizophrenia |
| ICD-10-CM DX | F325 | Major depressive disorder, single episode, in full remission |
| ICD-10-CM DX | F324 | Major depressive disorder, single episode, in partial remission |
| ICD-10-CM DX | F320 | Major depressive disorder, single episode, mild |
| ICD-10-CM DX | F321 | Major depressive disorder, single episode, moderate |
| ICD-10-CM DX | F323 | Major depressive disorder, single episode, severe with psychotic features |
| ICD-10-CM DX | F322 | Major depressive disorder, single episode, severe without psychotic features |
| ICD-10-CM DX | F25.x | Schizoaffective disorders |
| ICD-10-CM DX | F328 | Other specified depressive disorder |
| ICD-10-CM DX | F329 | Major depressive disorder, single episode, unspecified |
| ICD-10-CM DX | F332 | Major depressive disorder, recurrent severe without psychotic features |
| ICD-10-CM DX | F3342 | Major depressive disorder, recurrent, in full remission |
| ICD-10-CM DX | F3341 | Major depressive disorder, recurrent, in partial remission |
| ICD-10-CM DX | F3340 | Major depressive disorder, recurrent, in remission, unspecified |
| ICD-10-CM DX | F330 | Major depressive disorder, recurrent, mild |
| ICD-10-CM DX | F331 | Major depressive disorder, recurrent, moderate |
| ICD-10-CM DX | F333 | Major depressive disorder, recurrent, severe with psychotic symptoms |
| ICD-10-CM DX | F339 | Major depressive disorder, recurrent, unspecified |
| ICD-10-CM DX | F31.x | Manic depression/bipolar disorder |
| ICD-10-CM DX | F20.x | Schizophrenia |
| ICD-10-CM DX | F43.1 | Persistent depressive disorder |
| ICD-10-CM DX | F43.21 | Adjustment d/o with depressed mood |
| ICD-10-CM DX | F43.23 | Adjustment d/o with mixed anxiety and depressed mood |

| MEDICATION ID | NAME | GENERIC NAME | ORDER COUNT |
|---|---|---|---|
| 30792 | SERTRALINE HCL 50 MG PO TABS | Sertraline HCl Tab 50 MG | 364265 |
| 30792 | | Sertraline HCl Tab 30 MG Sertraline HCl Tab 100 MG | 344586 |
| 49150 | SERTRALINE HCL 100 MG PO TABS ESCITALOPRAM OXALATE 10 MG PO TABS | Escitalopram Oxalate Tab 10 MG (Base Equiv) | 279295 |
| 27521 | | Fluoxetine HCl Cap 20 MG | 250226 |
| 25473 | FLUOXETINE HCL 20 MG PO CAPS CITALOPRAM HYDROBROMIDE 20 MG PO TABS | Citalopram Hydrobromide Tab 20 MG (Base Equiv) | 246662 |
| 49151 | | Escitalopram Oxalate Tab 20 MG (Base Equiv) | 191759 |
| 52482 | BUPROPION HCL ER (XL) 150 MG PO TB24 | Bupropion HCl Tab ER 24HR 150 MG | 191739 |
| | BUPROPION NCL ER (AL) 130 MG PO 1B24 | Duloxetine HCl Enteric Coated Pellets Cap 60 MG (Base | 191323 |
| 54838 | DULOXETINE HCL 60 MG PO CPEP | Eq) | 179414 |
| 41375 | VENLAFAXINE HCL ER 75 MG PO CP24 | Venlafaxine HCl Cap ER 24HR 75 MG (Base Equivalent) Duloxetine HCl Enteric Coated Pellets Cap 30 MG (Base | 140523 |
| 54837 | DULOXETINE HCL 30 MG PO CPEP | Eq) | 140369 |
| 52483 | BUPROPION HCL ER (XL) 300 MG PO TB24 | Bupropion HCl Tab ER 24HR 300 MG | 136883 |
| 41377 | VENLAFAXINE HCL ER 150 MG PO CP24 | Venlafaxine HCl Cap ER 24HR 150 MG (Base Equivalent) | 129493 |
| 26233 | CITALOPRAM HYDROBROMIDE 40 MG PO TABS | Citalopram Hydrobromide Tab 40 MG (Base Equiv) | 128087 |
| 14668 | SERTRALINE HCL 25 MG PO TABS | Sertraline HCl Tab 25 MG | 126081 |
| 1130 | AMITRIPTYLINE HCL 25 MG PO TABS | Amitriptyline HCl Tab 25 MG | 111075 |
| 31120 | FLUOXETINE HCL 40 MG PO CAPS | Fluoxetine HCl Cap 40 MG | 110799 |
| 6802 | BUPROPION HCL ER (SR) 150 MG PO TB12 | Bupropion HCl Tab ER 12HR 150 MG | 110322 |
| 3069 | MIRTAZAPINE 15 MG PO TABS | Mirtazapine Tab 15 MG | 101445 |
| 29473 | PAROXETINE HCL 20 MG PO TABS | Paroxetine HCl Tab 20 MG | 93100 |
| 45710 | CITALOPRAM HYDROBROMIDE 10 MG PO TABS | Citalopram Hydrobromide Tab 10 MG (Base Equiv) | 88045 |
| 1127 | AMITRIPTYLINE HCL 10 MG PO TABS | Amitriptyline HCl Tab 10 MG | 84142 |
| 27520 | FLUOXETINE HCL 10 MG PO CAPS | Fluoxetine HCl Cap 10 MG | 76319 |
| | | Venlafaxine HCl Cap ER 24HR 37.5 MG (Base | |
| 41370 | VENLAFAXINE HCL ER 37.5 MG PO CP24 | Equivalent) | 64038 |
| 46525 | FLUOXETINE HCL 20 MG PO TABS | Fluoxetine HCl Tab 20 MG | 47822 |
| 43380 | PAROXETINE HCL 10 MG PO TABS | Paroxetine HCl Tab 10 MG | 46591 |
| 1131 | AMITRIPTYLINE HCL 50 MG PO TABS | Amitriptyline HCl Tab 50 MG | 42808 |
| 3068 | MIRTAZAPINE 30 MG PO TABS | Mirtazapine Tab 30 MG | 41887 |
| 43381 | PAROXETINE HCL 40 MG PO TABS | Paroxetine HCl Tab 40 MG | 41484 |
| 53289 | ESCITALOPRAM OXALATE 5 MG PO TABS | Escitalopram Oxalate Tab 5 MG (Base Equiv) | 40429 |
| 21941 | TRAZODONE HCL 150 MG PO TABS | Trazodone HCl Tab 150 MG | 40137 |
| 15185 | NORTRIPTYLINE HCL 10 MG PO CAPS | Nortriptyline HCl Cap 10 MG | 38909 |
| 33067 | VENLAFAXINE HCL 75 MG PO TABS | Venlafaxine HCl Tab 75 MG (Base Equivalent) | 35559 |
| 15186 | NORTRIPTYLINE HCL 25 MG PO CAPS | Nortriptyline HCl Cap 25 MG Duloxetine HCl Enteric Coated Pellets Cap 20 MG (Base | 33918 |
| 54836 | DULOXETINE HCL 20 MG PO CPEP | Eq) | 33170 |
| 49138 | LEXAPRO 10 MG PO TABS | Escitalopram Oxalate Tab 10 MG (Base Equiv) | 25964 |
| 29474 | PAROXETINE HCL 30 MG PO TABS | Paroxetine HCl Tab 30 MG | 25543 |
| 24234 | ZOLOFT 50 MG PO TABS | Sertraline HCl Tab 50 MG | 24619 |
| 6801 | BUPROPION HCL ER (SR) 100 MG PO TB12 | Bupropion HCl Tab ER 12HR 100 MG | 23869 |
| 54049 | MIRTAZAPINE 7.5 MG PO TABS | Mirtazapine Tab 7.5 MG | 23111 |
| 30269 | FLUOXETINE HCL 10 MG PO TABS | Fluoxetine HCl Tab 10 MG | 22273 |

| 25491 | BUPROPION HCL 75 MG PO TABS | Bupropion HCl Tab 75 MG | 21540 |
|---|---|---|---|
| 33068 | VENLAFAXINE HCL 37.5 MG PO TABS | Venlafaxine HCl Tab 37.5 MG (Base Equivalent) | 21070 |
| 24233 | ZOLOFT 100 MG PO TABS | Sertraline HCl Tab 100 MG | 20074 |
| 16385 | PAXIL 20 MG PO TABS | Paroxetine HCl Tab 20 MG | 18434 |
| 25490 | BUPROPION HCL 100 MG PO TABS | Bupropion HCl Tab 100 MG | 17921 |
| 18059 | PROZAC 20 MG PO CAPS | Fluoxetine HCl Cap 20 MG | 16426 |
| 7035 | DOXEPIN HCL 10 MG PO CAPS | Doxepin HCl Cap 10 MG | 16384 |
| 1128 | AMITRIPTYLINE HCL 100 MG PO TABS | Amitriptyline HCl Tab 100 MG | 16341 |
| | DESVENLAFAXINE SUCCINATE ER 50 MG PO | Desvenlafaxine Succinate Tab ER 24HR 50 MG (Base | |
| 72022 | TB24 | Equiv) | 15946 |
| 26237 | CELEXA 20 MG PO TABS | Citalopram Hydrobromide Tab 20 MG (Base Equiv) | 15281 |
| 15187 | NORTRIPTYLINE HCL 50 MG PO CAPS | Nortriptyline HCl Cap 50 MG | 14927 |
| 48727 | BUPROPION HCL ER (SR) 200 MG PO TB12 | Bupropion HCl Tab ER 12HR 200 MG | 14897 |
| 20977 | EFFEXOR XR 75 MG PO CP24 | Venlafaxine HCl Cap ER 24HR 75 MG (Base Equivalent) | 14669 |
| 29905 | MIRTAZAPINE 45 MG PO TABS | Mirtazapine Tab 45 MG | 12852 |
| 7038 | DOXEPIN HCL 25 MG PO CAPS | Doxepin HCl Cap 25 MG | 12040 |
| 49140 | LEXAPRO 20 MG PO TABS | Escitalopram Oxalate Tab 20 MG (Base Equiv) Duloxetine HCl Enteric Coated Pellets Cap 60 MG (Base | 10718 |
| 54830 | CYMBALTA 60 MG PO CPEP | Eq) | 10331 |
| 1132 | AMITRIPTYLINE HCL 75 MG PO TABS | Amitriptyline HCl Tab 75 MG | 9606 |
| 20979 | EFFEXOR XR 150 MG PO CP24 | Venlafaxine HCl Cap ER 24HR 150 MG (Base Equivalent) | 9586 |
| 72023 | DESVENLAFAXINE SUCCINATE ER 100 MG PO<br>TB24 | Desvenlafaxine Succinate Tab ER 24HR 100 MG (Base Equiv) | 9391 |
| 6825 | WELLBUTRIN SR 150 MG PO TBCR | NULL | 7725 |
| 7039 | DOXEPIN HCL 50 MG PO CAPS | Doxepin HCl Cap 50 MG | 7042 |
| 52480 | WELLBUTRIN XL 150 MG PO TB24 | Bupropion HCl Tab ER 24HR 150 MG | 6968 |
| 52481 | WELLBUTRIN XL 300 MG PO TB24 | Bupropion HCl Tab ER 24HR 300 MG | 6922 |
| 80523 | VILAZODONE HCL 40 MG PO TABS | Vilazodone HCl Tab 40 MG | 6849 |
| 43371 | PAXIL 10 MG PO TABS | Paroxetine HCl Tab 10 MG | 6813 |
| 44901 | MIRTAZAPINE 15 MG PO TBDP | Mirtazapine Orally Disintegrating Tab 15 MG | 6798 |
| 10582 | IMIPRAMINE HCL 25 MG PO TABS | Imipramine HCl Tab 25 MG | 6650 |
| 74599 | VENLAFAXINE HCL ER 150 MG PO TB24 | Venlafaxine HCl Tab ER 24HR 150 MG (Base Equivalent) | 6585 |
| 103956 | TRAZODONE HCL PO | traZODone HCl | 6562 |
| 54831 | CYMBALTA 30 MG PO CPEP | Duloxetine HCl Enteric Coated Pellets Cap 30 MG (Base Eq) | 6485 |
| 26238 | CELEXA 40 MG PO TABS | Citalopram Hydrobromide Tab 40 MG (Base Equiv) | 6402 |
| 27552 | FLUVOXAMINE MALEATE 100 MG PO TABS | Fluvoxamine Maleate Tab 100 MG | 6244 |
| 101719 | SERTRALINE HCL PO | Sertraline HCl | 5893 |
| 10583 | IMIPRAMINE HCL 50 MG PO TABS | Imipramine HCl Tab 50 MG | 5647 |
| 33064 | VENLAFAXINE HCL 25 MG PO TABS | Venlafaxine HCl Tab 25 MG (Base Equivalent) | 5629 |
| 33066 | VENLAFAXINE HCL 100 MG PO TABS | Venlafaxine HCl Tab 100 MG (Base Equivalent) | 5403 |
| 54119 | FLUOXETINE HCL 20 MG/5ML PO SOLN | Fluoxetine HCl Solution 20 MG/5ML | 4766 |
| 31386 | TRAZODONE HCL 300 MG PO TABS | Trazodone HCl Tab 300 MG | 4706 |
| 48243 | PAROXETINE HCL ER 25 MG PO TB24 | Paroxetine HCl Tab ER 24HR 25 MG | 4651 |
| 74598 | VENLAFAXINE HCL ER 75 MG PO TB24 | Venlafaxine HCl Tab ER 24HR 75 MG (Base Equivalent) | 4581 |

| 74600 | VENLAFAXINE HCL ER 225 MG PO TB24 | Venlafaxine HCl Tab ER 24HR 225 MG (Base Equivalent) | 4467 |
|---|---|---|---|
| 6241 | DESIPRAMINE HCL 25 MG PO TABS | Desipramine HCl Tab 25 MG | 4466 |
| 27553 | FLUVOXAMINE MALEATE 50 MG PO TABS | Fluvoxamine Maleate Tab 50 MG | 4418 |
| 20976 | EFFEXOR XR 37.5 MG PO CP24 | Venlafaxine HCl Cap ER 24HR 37.5 MG (Base Equivalent) | 4403 |
| 15188 | NORTRIPTYLINE HCL 75 MG PO CAPS | Nortriptyline HCl Cap 75 MG | 4326 |
| 52739 | WELLBUTRIN SR 150 MG PO TB12 | Bupropion HCl Tab ER 12HR 150 MG | 4203 |
| 12168 | ZOLOFT 25 MG PO TABS | Sertraline HCl Tab 25 MG | 4075 |
| 18058 | PROZAC 10 MG PO CAPS | Fluoxetine HCl Cap 10 MG | 3984 |
| 91500 | FLUOXETINE HCL PO | FLUoxetine HCl | 3908 |
| 37510 | EFFEXOR 75 MG PO TABS | Venlafaxine HCl Tab 75 MG (Base Equivalent) | 3893 |
| 43372 | PAXIL 40 MG PO TABS | Paroxetine HCl Tab 40 MG | 3812 |
| 87235 | CITALOPRAM HYDROBROMIDE PO | Citalopram Hydrobromide | 3777 |
| 105378 | WELLBUTRIN PO | buPROPion HCl | 3710 |
| 16386 | PAXIL 30 MG PO TABS | Paroxetine HCl Tab 30 MG | 3705 |
| 121792 | VORTIOXETINE HBR 10 MG PO TABS | Vortioxetine HBr Tab 10 MG (Base Equiv) | 3563 |
| 32736 | PROZAC 40 MG PO CAPS | Fluoxetine HCl Cap 40 MG | 3537 |
| 107520 | FLUOXETINE HCL 60 MG PO TABS | Fluoxetine HCl Tab 60 MG | 3446 |
| 80522 | VILAZODONE HCL 20 MG PO TABS | Vilazodone HCl Tab 20 MG | 3292 |
| 105801 | ZOLOFT PO | Sertraline HCl | 3283 |
| 33065 | VENLAFAXINE HCL 50 MG PO TABS | Venlafaxine HCl Tab 50 MG (Base Equivalent) | 3224 |
| 37994 | SERTRALINE HCL 20 MG/ML PO CONC | Sertraline HCl Oral Concentrate for Solution 20 MG/ML | 3209 |
| 1129 | AMITRIPTYLINE HCL 150 MG PO TABS | Amitriptyline HCl Tab 150 MG | 3202 |
| 48254 | PAXIL CR 25 MG PO TB24 | Paroxetine HCl Tab ER 24HR 25 MG | 3169 |
| 74597 | VENLAFAXINE HCL ER 37.5 MG PO TB24 | Venlafaxine HCl Tab ER 24HR 37.5 MG (Base Equivalent) | 3046 |
| 94580 | LEXAPRO PO | Escitalopram Oxalate | 2822 |
| 44902 | MIRTAZAPINE 30 MG PO TBDP | Mirtazapine Orally Disintegrating Tab 30 MG | 2795 |
| 7036 | DOXEPIN HCL 100 MG PO CAPS | Doxepin HCl Cap 100 MG | 2779 |
| 10581 | IMIPRAMINE HCL 10 MG PO TABS | Imipramine HCl Tab 10 MG | 2602 |
| 121793 | VORTIOXETINE HBR 20 MG PO TABS | Vortioxetine HBr Tab 20 MG (Base Equiv) | 2559 |
| 84163 | AMITRIPTYLINE HCL PO | Amitriptyline HCl | 2520 |
| 48242 | PAROXETINE HCL ER 12.5 MG PO TB24 | Paroxetine HCl Tab ER 24HR 12.5 MG | 2485 |
| 86048 | BUPROPION HCL PO | buPROPion HCl | 2454 |
| 48253 | PAXIL CR 12.5 MG PO TB24 | Paroxetine HCl Tab ER 24HR 12.5 MG | 2367 |
| 88576 | CYMBALTA PO | DULoxetine HCl | 2273 |
| 4753 | CLOMIPRAMINE HCL 50 MG PO CAPS | Clomipramine HCl Cap 50 MG | 2260 |
| 99459 | PROZAC PO | FLUoxetine HCl | 2168 |
| 45716 | CELEXA 10 MG PO TABS | Citalopram Hydrobromide Tab 10 MG (Base Equiv) | 2162 |
| 48244 | PAROXETINE HCL ER 37.5 MG PO TB24 | Paroxetine HCl Tab ER 24HR 37.5 MG | 2150 |
| 128150 | DESVENLAFAXINE SUCCINATE ER 25 MG PO<br>TB24 | Desvenlafaxine Succinate Tab ER 24HR 25 MG (Base Equiv) | 1978 |
| 115687 | BUPROPION HCL ER (XL) 450 MG PO TB24 | Bupropion HCl Tab ER 24HR 450 MG | 1965 |
| 72176 | PRISTIQ 50 MG PO TB24 | Desvenlafaxine Succinate Tab ER 24HR 50 MG (Base Equiv) | 1951 |
| 37511 | EFFEXOR 37.5 MG PO TABS | Venlafaxine HCl Tab 37.5 MG (Base Equivalent) | 1899 |

| 128921 | DULOXETINE HCL 40 MG PO CPEP | Duloxetine HCl Enteric Coated Pellets Cap 40 MG (Base Eq) | 1710 |
|---|---|---|---|
| 44894 | REMERON SOLTAB 30 MG PO TBDP | Mirtazapine Orally Disintegrating Tab 30 MG | 1696 |
| 26357 | CLOMIPRAMINE HCL 25 MG PO CAPS | Clomipramine HCl Cap 25 MG | 1674 |
| 6242 | DESIPRAMINE HCL 50 MG PO TABS | Desipramine HCl Tab 50 MG | 1638 |
| 3093 | REMERON 15 MG PO TABS | Mirtazapine Tab 15 MG | 1593 |
| 80521 | VILAZODONE HCL 10 MG PO TABS | Vilazodone HCl Tab 10 MG | 1563 |
| 44893 | REMERON SOLTAB 15 MG PO TBDP | Mirtazapine Orally Disintegrating Tab 15 MG | 1518 |
| 7491 | ELAVIL 25 MG PO TABS | Amitriptyline HCl Tab 25 MG | 1500 |
| 7488 | ELAVIL 10 MG PO TABS | Amitriptyline HCl Tab 10 MG | 1450 |
| 7040 | DOXEPIN HCL 75 MG PO CAPS | Doxepin HCl Cap 75 MG | 1436 |
| 3094 | REMERON 30 MG PO TABS | Mirtazapine Tab 30 MG | 1391 |
| 6823 | WELLBUTRIN SR 100 MG PO TBCR | NULL | 1388 |
| 6238 | DESIPRAMINE HCL 10 MG PO TABS | Desipramine HCl Tab 10 MG | 1360 |
| 72177 | PRISTIQ 100 MG PO TB24 | Desvenlafaxine Succinate Tab ER 24HR 100 MG (Base Equiv) | 1336 |
| | | Duloxetine HCl Enteric Coated Pellets Cap 20 MG (Base | |
| 54829 | CYMBALTA 20 MG PO CPEP | Eq) | 1308 |
| 90158 | EFFEXOR PO | Venlafaxine HCl | 1307 |
| 23872 | WELLBUTRIN 100 MG PO TABS | Bupropion HCl Tab 100 MG | 1266 |
| 104831 | VENLAFAXINE HCL PO | Venlafaxine HCl | 1255 |
| 53337 | LEXAPRO 5 MG PO TABS | Escitalopram Oxalate Tab 5 MG (Base Equiv) | 1189 |
| 80922 | VIIBRYD 40 MG PO TABS | Vilazodone HCl Tab 40 MG | 1167 |
| 36044 | NEFAZODONE HCL 100 MG PO TABS | Nefazodone HCl Tab 100 MG<br>Levomilnacipran HCl Cap ER 24HR 40 MG (Base | 1121 |
| 122218 | LEVOMILNACIPRAN HCL ER 40 MG PO CP24 | Equivalent) | 1079 |
| 90794 | ESCITALOPRAM OXALATE PO CITALOPRAM HYDROBROMIDE 10 MG/5ML PO | Escitalopram Oxalate | 1059 |
| 38018 | SOLN SOLN | Citalopram Hydrobromide Oral Soln 10 MG/5ML | 1041 |
| 50590 | ESCITALOPRAM OXALATE 5 MG/5ML PO SOLN | Escitalopram Oxalate Soln 5 MG/5ML (Base Equiv) | 1022 |
| 36046 | NEFAZODONE HCL 200 MG PO TABS | Nefazodone HCl Tab 200 MG | 982 |
| 36045 | NEFAZODONE HCL 150 MG PO TABS | Nefazodone HCl Tab 150 MG | 977 |
| 17917 | FLUVOXAMINE MALEATE 25 MG PO TABS | Fluvoxamine Maleate Tab 25 MG | 965 |
| 89706 | DULOXETINE HCL PO | DULoxetine HCl | 940 |
| 7037 | DOXEPIN HCL 150 MG PO CAPS | Doxepin HCl Cap 150 MG | 929 |
| 97999 | PAXIL PO | PARoxetine HCl | 913 |
| 26358 | CLOMIPRAMINE HCL 75 MG PO CAPS | Clomipramine HCl Cap 75 MG | 911 |
| 23873 | WELLBUTRIN 75 MG PO TABS | Bupropion HCl Tab 75 MG | 875 |
| 30321 | PROTRIPTYLINE HCL 5 MG PO TABS | Protriptyline HCl Tab 5 MG | 860 |
| 97988 | PAROXETINE HCL PO | PARoxetine HCl | 852 |
| 38229 | SERZONE 150 MG PO TABS | Nefazodone HCl Tab 150 MG | 837 |
| 30320 | PROTRIPTYLINE HCL 10 MG PO TABS | Protriptyline HCl Tab 10 MG | 828 |
| 95905 | MIRTAZAPINE PO | Mirtazapine | 820 |
| 121791 | VORTIOXETINE HBR 5 MG PO TABS | Vortioxetine HBr Tab 5 MG (Base Equiv) | 817 |
| 52738 | WELLBUTRIN SR 100 MG PO TB12 | Bupropion HCl Tab ER 12HR 100 MG | 804 |
| 72073 | FLUVOXAMINE MALEATE ER 100 MG PO CP24 | Fluvoxamine Maleate Cap ER 24HR 100 MG | 764 |

| 122219 | LEVOMILNACIPRAN HCL ER 80 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 80 MG (Base Equivalent) | 764 |
|---|---|---|---|
| 86679 | CELEXA PO | Citalopram Hydrobromide | 752 |
| 48255 | PAXIL CR 37.5 MG PO TB24 | Paroxetine HCl Tab ER 24HR 37.5 MG | 740 |
| 52740 | WELLBUTRIN SR 200 MG PO TB12 | Bupropion HCl Tab ER 12HR 200 MG | 712 |
| 45394 | MIRTAZAPINE 45 MG PO TBDP | Mirtazapine Orally Disintegrating Tab 45 MG | 695 |
| 38228 | SERZONE 200 MG PO TABS | Nefazodone HCl Tab 200 MG | 661 |
| 45212 | PROZAC WEEKLY 90 MG PO CPDR | Fluoxetine HCl Cap Delayed Release 90 MG | 653 |
| 90159 | EFFEXOR XR PO | Venlafaxine HCl | 653 |
| 113119 | VILAZODONE HCL 10 & 20 & 40 MG PO KIT | Vilazodone HCl Tab Starter Kit 10 (7) & 20 (7) & 40 (16) | 620 |
| 122220 | LEVOMILNACIPRAN HCL ER 120 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 120 MG (Base Equivalent) | 596 |
| 38227 | SERZONE 100 MG PO TABS | Nefazodone HCl Tab 100 MG | 589 |
| 45213 | FLUOXETINE HCL 90 MG PO CPDR | Fluoxetine HCl Cap Delayed Release 90 MG | 561 |
| 72074 | FLUVOXAMINE MALEATE ER 150 MG PO CP24 | Fluvoxamine Maleate Cap ER 24HR 150 MG | 553 |
| 122217 | LEVOMILNACIPRAN HCL ER 20 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 20 MG (Base Equivalent) | 547 |
| 29910 | REMERON 45 MG PO TABS | Mirtazapine Tab 45 MG | 526 |
| 6239 | DESIPRAMINE HCL 100 MG PO TABS | Desipramine HCl Tab 100 MG | 510 |
| 7041 | DOXEPIN HCL 10 MG/ML PO CONC | Doxepin HCl Cone 10 MG/ML | 495 |
| 29648 | PHENELZINE SULFATE 15 MG PO TABS | Phenelzine Sulfate Tab 15 MG | 487 |
| 7492 | ELAVIL 50 MG PO TABS | Amitriptyline HCl Tab 50 MG | 469 |
| 119146 | DESVENLAFAXINE ER 50 MG PO TB24 | Desvenlafaxine Tab ER 24HR 50 MG | 465 |
| 97070 | NORTRIPTYLINE HCL PO | Nortriptyline HCl | 439 |
| 82218 | TRAZODONE HCL ER 150 MG PO TB24 | Trazodone HCl Tab ER 24HR 150 MG | 431 |
| 37509 | EFFEXOR 100 MG PO TABS | Venlafaxine HCl Tab 100 MG (Base Equivalent) | 430 |
| 29178 | NORTRIPTYLINE HCL 10 MG/5ML PO SOLN | Nortriptyline HCl Soln 10 MG/5ML | 410 |
| 99177 | PRISTIQ PO | Desvenlafaxine Succinate | 404 |
| 24605 | PAROXETINE HCL 10 MG/5ML PO SUSP | Paroxetine HCl Oral Susp 10 MG/5ML (Base Equiv) | 401 |
| 48739 | WELLBUTRIN SR 200 MG PO TBCR | NULL | 379 |
| 132523 | TRINTELLIX 20 MG PO TABS | Vortioxetine HBr Tab 20 MG (Base Equiv) | 361 |
| 30290 | PROZAC 10 MG PO TABS | Fluoxetine HCl Tab 10 MG | 358 |
| 105380 | WELLBUTRIN XL PO | buPROPion HCl | 343 |
| 80921 | VIIBRYD 20 MG PO TABS | Vilazodone HCl Tab 20 MG | 338 |
| 6243 | DESIPRAMINE HCL 75 MG PO TABS | Desipramine HCl Tab 75 MG | 337 |
| 100750 | REMERON PO | Mirtazapine | 336 |
| 132522 | TRINTELLIX 10 MG PO TABS | Vortioxetine HBr Tab 10 MG (Base Equiv) | 324 |
| 37507 | EFFEXOR 25 MG PO TABS | Venlafaxine HCl Tab 25 MG (Base Equivalent) | 311 |
| 119147 | DESVENLAFAXINE ER 100 MG PO TB24 | Desvenlafaxine Tab ER 24HR 100 MG | 283 |
| 19392 | NEFAZODONE HCL 50 MG PO TABS | Nefazodone HCl Tab 50 MG | 269 |
| 82549 | VIIBRYD PO | Vilazodone HCl | 266 |
| 53826 | BUDEPRION SR 150 MG PO TB12 | Bupropion HCl Tab ER 12HR 150 MG | 263 |
| 37508 | EFFEXOR 50 MG PO TABS | Venlafaxine HCl Tab 50 MG (Base Equivalent) | 258 |
| 27929 | IMIPRAMINE PAMOATE 75 MG PO CAPS | Imipramine Pamoate Cap 75 MG | 245 |
| 27926 | IMIPRAMINE PAMOATE 100 MG PO CAPS | Imipramine Pamoate Cap 100 MG | 238 |

| 23796 | VIVACTIL 10 MG PO TABS | Protriptyline HCl Tab 10 MG | 235 |
|---|---|---|---|
| 1156 | AMOXAPINE 50 MG PO TABS | Amoxapine Tab 50 MG | 235 |
| 37925 | LUVOX 100 MG PO TABS | Fluvoxamine Maleate Tab 100 MG | 228 |
| 16153 | PAMELOR 10 MG PO CAPS | Nortriptyline HCl Cap 10 MG | 226 |
| 89586 | DOXEPIN HCL PO | Doxepin HCl | 225 |
| 53112 | PAROXETINE MESYLATE 20 MG PO TABS | Paroxetine Mesylate Tab 20 MG (Base Equiv) | 221 |
| 31385 | TRANYLCYPROMINE SULFATE 10 MG PO TABS | Tranylcypromine Sulfate Tab 10 MG | 216 |
| 129677 | VILAZODONE HCL 10 & 20 MG PO KIT | Vilazodone HCl Tab Starter Kit 10 (7) & 20 (23) MG | 203 |
| 7493 | ELAVIL 75 MG PO TABS | Amitriptyline HCl Tab 75 MG | 197 |
| 1153 | AMOXAPINE 100 MG PO TABS | Amoxapine Tab 100 MG | 195 |
| 61428 | BUDEPRION XL 300 MG PO TB24 | Bupropion HCl Tab ER 24HR 300 MG | 192 |
| 122246 | LEVOMILNACIPRAN HCL ER 20 & 40 MG PO<br>C4PK | Levomilnacipran HCl Cap ER 24HR 20 & 40 MG<br>Therapy Pack | 192 |
| 19852 | SERZONE 50 MG PO TABS | Nefazodone HCl Tab 50 MG | 183 |
| 1155 | AMOXAPINE 25 MG PO TABS | Amoxapine Tab 25 MG | 183 |
| 72990 | BUDEPRION XL 150 MG PO TB24 | Bupropion HCl Tab ER 24HR 150 MG | 181 |
| 59776 | SELEGILINE 6 MG/24HR TD PT24 | Selegiline TD Patch 24HR 6 MG/24HR | 175 |
| 38259 | NEFAZODONE HCL 250 MG PO TABS | Nefazodone HCl Tab 250 MG | 157 |
| 16154 | PAMELOR 25 MG PO CAPS | Nortriptyline HCl Cap 25 MG | 156 |
| 37926 | LUVOX 50 MG PO TABS | Fluvoxamine Maleate Tab 50 MG | 150 |
| 7489 | ELAVIL 100 MG PO TABS | Amitriptyline HCl Tab 100 MG | 146 |
| 103953 | TRAZAMINE PO | NULL | 143 |
| 132712 | TRINTELLIX PO | Vortioxetine HBr | 141 |
| 122242 | FETZIMA 80 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 80 MG (Base Equivalent) | 138 |
| 12816 | MAPROTILINE HCL 50 MG PO TABS | Maprotiline HCl Tab 50 MG | 138 |
| 27928 | IMIPRAMINE PAMOATE 150 MG PO CAPS | Imipramine Pamoate Cap 150 MG | 134 |
| 6240 | DESIPRAMINE HCL 150 MG PO TABS | Desipramine HCl Tab 150 MG | 134 |
| 80920 | VIIBRYD 10 MG PO TABS | Vilazodone HCl Tab 10 MG | 126 |
| 53114 | PAROXETINE MESYLATE 40 MG PO TABS | Paroxetine Mesylate Tab 40 MG (Base Equiv) | 124 |
| 24603 | PAXIL 10 MG/5ML PO SUSP | Paroxetine HCl Oral Susp 10 MG/5ML (Base Equiv) | 122 |
| 115898 | FORFIVO XL 450 MG PO TB24 | Bupropion HCl Tab ER 24HR 450 MG | 122 |
| 45380 | REMERON SOLTAB 45 MG PO TBDP | Mirtazapine Orally Disintegrating Tab 45 MG | 117 |
| 53111 | PAROXETINE MESYLATE 10 MG PO TABS | Paroxetine Mesylate Tab 10 MG (Base Equiv) | 117 |
| 1230 | ANAFRANIL 50 MG PO CAPS | Clomipramine HCl Cap 50 MG | 112 |
| 122245 | FETZIMA 40 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 40 MG (Base Equivalent) | 109 |
| 12815 | MAPROTILINE HCL 25 MG PO TABS | Maprotiline HCl Tab 25 MG | 106 |
| 16155 | PAMELOR 50 MG PO CAPS | Nortriptyline HCl Cap 50 MG | 105 |
| 59778 | SELEGILINE 12 MG/24HR TD PT24 | Selegiline TD Patch 24HR 12 MG/24HR | 103 |
| 116927 | BUPROPION HBR ER PO | buPROPion HBr | 99 |
| 97071 | NORTRIPYTLINE HCL PO | Nortriptyline HCl | 93 |
| 122243 | FETZIMA 120 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 120 MG (Base Equivalent) | 92 |
| 105379 | WELLBUTRIN SR PO | buPROPion HCl | 89 |
| 38230 | SERZONE 250 MG PO TABS | Nefazodone HCl Tab 250 MG | 86 |

| 14441 | NARDIL 15 MG PO TABS | Phenelzine Sulfate Tab 15 MG | 82 |
|---|---|---|---|
| 117245 | VENLAFAXINE HCL ER PO | Venlafaxine HCl | 82 |
| 86043 | BUPROPION HBR PO | buPROPion HBr | 80 |
| 20758 | SURMONTIL 50 MG PO CAPS | Trimipramine Maleate Cap 50 MG | 78 |
| 38025 | CELEXA 10 MG/5ML PO SOLN | Citalopram Hydrobromide Oral Soln 10 MG/5ML | 78 |
| 37993 | ZOLOFT 20 MG/ML PO CONC | Sertraline HCl Oral Concentrate for Solution 20 MG/ML | 74 |
| 116013 | BUPROPION HCL ER (SR) PO | buPROPion HCl | 74 |
| 53113 | PAROXETINE MESYLATE 30 MG PO TABS | Paroxetine Mesylate Tab 30 MG (Base Equiv) | 73 |
| 53251 | PEXEVA 20 MG PO TABS | Paroxetine Mesylate Tab 20 MG (Base Equiv) | 71 |
| 59777 | SELEGILINE 9 MG/24HR TD PT24 | Selegiline TD Patch 24HR 9 MG/24HR | 70 |
| 1229 | ANAFRANIL 25 MG PO CAPS | Clomipramine HCl Cap 25 MG | 69 |
| 21746 | TOFRANIL 25 MG PO TABS | Imipramine HCl Tab 25 MG | 69 |
| 75930 | BUPROPION HBR ER 522 MG PO TB24 | Bupropion HBr Tab ER 24HR 522 MG | 66 |
| 82219 | TRAZODONE HCL ER 300 MG PO TB24 | Trazodone HCl Tab ER 24HR 300 MG | 66 |
| 93521 | IMIPRAMINE HCL PO | Imipramine HCl | 64 |
| 132521 | TRINTELLIX 5 MG PO TABS | Vortioxetine HBr Tab 5 MG (Base Equiv) | 63 |
| 122496 | FETZIMA PO | Levomilnacipran HCl | 61 |
| 116014 | BUPROPION HCL ER (XL) PO | buPROPion HCl | 60 |
| 21747 | TOFRANIL 50 MG PO TABS | Imipramine HCl Tab 50 MG | 58 |
| 400628 | VENLAFAXINE(COMPOUNDED) 15 MG/ML PO<br>SUSP | venlafaxine (compounded) 15 mg/mL po susp | 57 |
| 117239 | TRAZODONE HCL ER PO | traZODone HCl | 55 |
| 6271 | DESYREL 150 MG PO TABS | Trazodone HCl Tab 150 MG | 54 |
| 1154 | AMOXAPINE 150 MG PO TABS | Amoxapine Tab 150 MG | 53 |
| 15182 | NORPRAMIN 25 MG PO TABS | Desipramine HCl Tab 25 MG | 53 |
| 95046 | LUVOX CR PO | fluvoxaMINE Maleate | 53 |
| 12817 | MAPROTILINE HCL 75 MG PO TABS | Maprotiline HCl Tab 75 MG | 51 |
| 55184 | PROZAC 20 MG/5ML PO SOLN | Fluoxetine HCl Solution 20 MG/5ML | 49 |
| 75223 | CITALOPRAM & DIET MANAGE PROD 10 MG PO<br>MISC | Citalopram Tab 10 MG & Dietary Management Cap Pack | 47 |
| 32005 | NORTRIPYTLINE HCL 25 MG PO CAPS | Nortriptyline HCl Cap 25 MG | 47 |
| 121979 | BRINTELLIX PO | Vortioxetine HBr | 46 |
| 87415 | CLOMIPRAMINE HCL PO | clomiPRAMINE HCl | 46 |
| 128151 | PRISTIQ 25 MG PO TB24 | Desvenlafaxine Succinate Tab ER 24HR 25 MG (Base Equiv) | 45 |
| 72075 | LUVOX CR 100 MG PO CP24 | Fluvoxamine Maleate Cap ER 24HR 100 MG | 45 |
| 15737 | LUVOX 25 MG PO TABS | Fluvoxamine Maleate Tab 25 MG | 43 |
| 91526 | FLUVOXAMINE MALEATE PO | fluvoxaMINE Maleate | 43 |
| 122244 | FETZIMA 20 MG PO CP24 | Levomilnacipran HCl Cap ER 24HR 20 MG (Base Equivalent) | 42 |
| 76881 | BUPROPION HBR ER 174 MG PO TB24 | Bupropion HBr Tab ER 24HR 174 MG | 41 |
| 6272 | DESYREL 300 MG PO TABS | Trazodone HCl Tab 300 MG | 41 |
| 18060 | PROZAC 20 MG/5ML PO LIQD | NULL | 38 |
| 132397 | ELAVIL PO | Amitriptyline HCl | 37 |
| 123813 | DESVENLAFAXINE FUMARATE ER 50 MG PO<br>TB24 | Desvenlafaxine Fumarate Tab ER 24HR 50 MG (Base Equiv) | 33 |
| 143013 | FLUOXETINE HCL 20 MG/5ML PO LIQD | NULL | 33 |

| 2057 | TRAZODONE HCL POWD | Trazodone HCl Powder | 33 |
|---|---|---|---|
| 1126 | AMITRIPTYLINE HCL 10 MG/ML IM SOLN | NULL | 33 |
| 75929 | BUPROPION HBR ER 348 MG PO TB24 | Bupropion HBr Tab ER 24HR 348 MG | 32 |
| 22238 | TRIMIPRAMINE MALEATE 25 MG PO CAPS | Trimipramine Maleate Cap 25 MG | 32 |
| 22239 | TRIMIPRAMINE MALEATE 50 MG PO CAPS | Trimipramine Maleate Cap 50 MG | 32 |
| 16156 | PAMELOR 75 MG PO CAPS | Nortriptyline HCl Cap 75 MG | 32 |
| 7490 | ELAVIL 150 MG PO TABS | Amitriptyline HCl Tab 150 MG | 32 |
| 72076 | LUVOX CR 150 MG PO CP24 | Fluvoxamine Maleate Cap ER 24HR 150 MG | 31 |
| 22237 | TRIMIPRAMINE MALEATE 100 MG PO CAPS | Trimipramine Maleate Cap 100 MG | 30 |
| 19544 | SINEQUAN 50 MG PO CAPS | Doxepin HCl Cap 50 MG | 29 |
| 50589 | LEXAPRO 5 MG/5ML PO SOLN | Escitalopram Oxalate Soln 5 MG/5ML (Base Equiv) | 29 |
| 119271 | DESVENLAFAXINE ER PO | Desvenlafaxine | 27 |
| 27927 | IMIPRAMINE PAMOATE 125 MG PO CAPS | Imipramine Pamoate Cap 125 MG | 27 |
| 121840 | BRINTELLIX 10 MG PO TABS | Vortioxetine HBr Tab 10 MG (Base Equiv) | 27 |
| 121841 | BRINTELLIX 20 MG PO TABS | Vortioxetine HBr Tab 20 MG (Base Equiv) | 27 |
| 96617 | NEFAZODONE HCL PO | Nefazodone HCl | 26 |
| 53253 | PEXEVA 40 MG PO TABS | Paroxetine Mesylate Tab 40 MG (Base Equiv) | 26 |
| 82550 | VILAZODONE HCL PO | Vilazodone HCl | 26 |
| 19545 | SINEQUAN 75 MG PO CAPS | Doxepin HCl Cap 75 MG | 25 |
| 97998 | PAXIL CR PO | PARoxetine HCl | 24 |
| 23797 | VIVACTIL 5 MG PO TABS | Protriptyline HCl Tab 5 MG | 22 |
| 89055 | DESYREL PO | traZODone HCl | 21 |
| 97989 | PAROXETINE MESYLATE PO | PARoxetine Mesylate | 20 |
| 53633 | BUDEPRION SR 100 MG PO TB12 | Bupropion HCl Tab ER 12HR 100 MG | 20 |
| 53252 | PEXEVA 30 MG PO TABS | Paroxetine Mesylate Tab 30 MG (Base Equiv) | 19 |
| 59804 | EMSAM 6 MG/24HR TD PT24 | Selegiline TD Patch 24HR 6 MG/24HR | 19 |
| 89011 | DESIPRAMINE HCL PO | Desipramine HCl | 19 |
| 113548 | VIIBRYD 10 & 20 & 40 MG PO KIT | Vilazodone HCl Tab Starter Kit 10 (7) & 20 (7) & 40 (16) MG | 19 |
| 84224 | ANAFRANIL PO | clomiPRAMINE HCl | 18 |
| 76061 | APLENZIN 522 MG PO TB24 | Bupropion HBr Tab ER 24HR 522 MG | 18 |
| 20756 | SURMONTIL 100 MG PO CAPS | Trimipramine Maleate Cap 100 MG | 18 |
| 20757 | SURMONTIL 25 MG PO CAPS | Trimipramine Maleate Cap 25 MG | 17 |
| 53250 | PEXEVA 10 MG PO TABS | Paroxetine Mesylate Tab 10 MG (Base Equiv) | 17 |
| 123815 | DESVENLAFAXINE FUMARATE ER 100 MG PO<br>TB24 | Desvenlafaxine Fumarate Tab ER 24HR 100 MG (Base Equiv) | 17 |
| 99446 | PROTRIPTYLINE HCL PO | Protriptyline HCl | 17 |
| 116975 | DESVENLAFAXINE SUCCINATE ER PO | Desvenlafaxine Succinate | 16 |
| 97884 | PAMELOR PO | Nortriptyline HCl | 15 |
| 1231 | ANAFRANIL 75 MG PO CAPS | Clomipramine HCl Cap 75 MG | 15 |
| 21751 | TOFRANIL-PM 75 MG PO CAPS | Imipramine Pamoate Cap 75 MG | 15 |
| 122259 | FETZIMA TITRATION 20 & 40 MG PO C4PK | Levomilnacipran HCl Cap ER 24HR 20 & 40 MG<br>Therapy Pack | 14 |
| 16338 | PARNATE 10 MG PO TABS | Tranylcypromine Sulfate Tab 10 MG | 14 |
| 129681 | VIIBRYD STARTER PACK 10 & 20 MG PO KIT | Vilazodone HCl Tab Starter Kit 10 (7) & 20 (23) MG | 14 |

| 87234 | CITALOPRAM & DIET MANAGE PROD PO | NULL | 12 |
|---|---|---|---|
| 19541 | SINEQUAN 100 MG PO CAPS | Doxepin HCl Cap 100 MG | 12 |
| 59874 | EMSAM 12 MG/24HR TD PT24 | Selegiline TD Patch 24HR 12 MG/24HR | 11 |
| 103954 | TRAZODONE & DIET MANAGE PROD PO | NULL | 10 |
| 76060 | APLENZIN 348 MG PO TB24 | Bupropion HBr Tab ER 24HR 348 MG | 10 |
| 15183 | NORPRAMIN 50 MG PO TABS | Desipramine HCl Tab 50 MG | 10 |
| 15179 | NORPRAMIN 30 MG PO TABS | Desipramine HCl Tab 10 MG | 10 |
| 19543 | | | 10 |
| 84189 | SINEQUAN 25 MG PO CAPS | Doxepin HCl Cap 25 MG Amoxapine | 9 |
| | AMOXAPINE PO | | 8 |
| 21745 | TOFRANIL 10 MG PO TABS | Imipramine HCl Tab 10 MG | 8 |
| 96477<br>68121 | NARDIL PO FLUOXETINE & DIET MANAGE PROD 10 MG PO MISC | Phenelzine Sulfate Fluoxetine HCl Cap 10 MG & Dietary Management Cap Pack | 8 |
| 59871 | EMSAM 9 MG/24HR TD PT24 | Selegiline TD Patch 24HR 9 MG/24HR | 7 |
| 1891 | ASENDIN TABS 50 MG PO | Amoxapine Tab 50 MG | 7 |
| 98330 | PEXEVA PO | PARoxetine Mesylate | 7 |
| 19540 | SINEOUAN 10 MG PO CAPS | Doxepin HCl Cap 10 MG | 7 |
| 108627 | BUPROPION HCL (XL) PO | buPROPion HCl | 7 |
| 117143 | PAROXETINE HCL ER PO | PARoxetine HCl | 6 |
| 108626 | BUPROPION HCL (SR) PO | buPROPion HCl | 6 |
| 15180 | NORPRAMIN 100 MG PO TABS | Desipramine HCl Tab 100 MG | 6 |
| 7487 | | NULL | 6 |
| 27338 | ELAVIL 10 MG/ML IM SOLN ISOCARBOXAZID 10 MG PO TABS | Isocarboxazid Tab 10 MG | 6 |
| 97986 | PARNATE PO | Tranylcypromine Sulfate | 5 |
| 85979 | BUDEPRION XL PO | buPROPion HCl | 5 |
| 85978 | BUDEPRION SR PO | buPROPion HCl | 5 |
| 63976 | AMITRIPTYLINE & DIET MANAGE PR 25 MG PO | Amitriptyline HCl Tab 25 MG & Diet Manage Prod Cap | 3 |
| 75165 | MISC | Pack | 5 |
| 105240 | VIVACTIL PO | Protriptyline HCl | 5 |
| 84461 | APLENZIN PO | buPROPion HBr | 5 |
| 122087 | VORTIOXETINE HBR PO | Vortioxetine HBr | 5 |
| 99460 | PROZAC WEEKLY PO | FLUoxetine HCl | 4 |
| 130049 | VIIBRYD STARTER PACK PO | Vilazodone HCl | 4 |
| 103824 | TOFRANIL PO | Imipramine HCl | 4 |
| 117032 | FLUVOXAMINE MALEATE ER PO | fluvoxaMINE Maleate | 4 |
| 21750 | TOFRANIL-PM 150 MG PO CAPS | Imipramine Pamoate Cap 150 MG | 4 |
| 98385 | PHENELZINE SULFATE PO | Phenelzine Sulfate | 4 |
| 16157 | PAMELOR 10 MG/5ML PO SOLN | Nortriptyline HCl Soln 10 MG/5ML | 4 |
| 19542 | SINEQUAN 150 MG PO CAPS | Doxepin HCl Cap 150 MG | 3 |
| 21749 | TOFRANIL-PM 125 MG PO CAPS | Imipramine Pamoate Cap 125 MG | 3 |
| 104125 | TRIMIPRAMINE MALEATE PO | Trimipramine Maleate | 3 |
| 97063 | NORPRAMIN PO | Desipramine HCl | 3 |
| 103921 | TRANYLCYPROMINE SULFATE PO | Tranylcypromine Sulfate | 3 |
| 2099 | NORTRIPTYLINE HCL POWD | Nortriptyline HCl Powder | 3 |

| 148925 | ESKETAMINE HCL (56 MG DOSE) 28 MG/DEVICE<br>NA SOPK | Esketamine HCl Nasal Soln 28 MG/Device x 2 (56 MG Dose Pack) | 3 |
|---|---|---|---|
| 100571 | RAPIFLUX PO | FLUoxetine HCl | 3 |
| 86042 | BUPROPION & DIET MANAGE PROD PO | NULL | 3 |
| 91770 | GABOXETINE PO | NULL | 3 |
| 91498 | FLUOXETINE & DIET MANAGE PROD PO | NULL | 3 |
| 90276 | EMSAM TD | Selegiline | 2 |
| 82404 | OLEPTRO 300 MG PO TB24 | Trazodone HCl Tab ER 24HR 300 MG | 2 |
| 82403 | OLEPTRO 150 MG PO TB24 | Trazodone HCl Tab ER 24HR 150 MG | 2 |
| 100751 | REMERON SOLTAB PO | Mirtazapine | 2 |
| 93522 | IMIPRAMINE PAMOATE PO | Imipramine Pamoate | 2 |
| 95225 | MAPROTILINE HCL PO | Maprotiline HCl | 2 |
| 121507 | KHEDEZLA PO | Desvenlafaxine | 2 |
| 148927 | ESKETAMINE HCL (84 MG DOSE) 28 MG/DEVICE<br>NA SOPK | Esketamine HCl Nasal Soln 28 MG/Device x 3 (84 MG Dose Pack) | 2 |
| 1881 | IMIPRAMINE HCL POWD | Imipramine HCl Powder | 2 |
| 68122 | GABOXETINE 10 MG PO MISC | Fluoxetine HCl Cap 10 MG & Dietary Management Cap<br>Pack | 2 |
| 21748 | TOFRANIL-PM 100 MG PO CAPS | Imipramine Pamoate Cap 100 MG | 2 |
| 27248 | MARPLAN 10 MG PO TABS | Isocarboxazid Tab 10 MG | 2 |
| 15181 | NORPRAMIN 150 MG PO TABS | Desipramine HCl Tab 150 MG | 1 |
| 103825 | TOFRANIL-PM PO | Imipramine Pamoate | 1 |
| 116112 | FORFIVO XL PO | buPROPion HCl | 1 |
| 97358 | OLEPTRO PO | traZODone HCl | 1 |
| 149210 | SPRAVATO (84 MG DOSE) NA | Esketamine HCl | 1 |
| 121369 | KHEDEZLA 100 MG PO TB24 | Desvenlafaxine Tab ER 24HR 100 MG | 1 |
| 121368 | KHEDEZLA 50 MG PO TB24 | Desvenlafaxine Tab ER 24HR 50 MG | 1 |
| 121839 | BRINTELLIX 5 MG PO TABS | Vortioxetine HBr Tab 5 MG (Base Equiv) | 1 |
| 101698 | SENTRAVIL PM-25 PO | NULL | 1 |
| 89054 | DESVENLAFAXINE SUCCINATE PO | Desvenlafaxine Succinate | 1 |

Notes: Trazodone less than 150mg, Amitriptyline, Nortriptyline, Imipramine, and Amoxapine may be excluded. NULL = Medication record is not linked to Generic Name.

| Appendix 3: ICD codes to identify patients with comorbidities | | |
|---|---|---|
| Code Type | Code or Code Range | Condition |
| ICD-9-CM DX | 3310 | Alzheimer's |
| ICD-10-CM DX | G30.x | Alzheimer's |
| ICD-9-CM DX | 14.x- 209.x | Cancer |
| ICD-10-CM DX | C0.x-C96.x | Cancer |
| ICD-9-CM DX | 43.x-44.39; 7854, V434 | Cerebrovascular |
| | | disease |
| ICD-10-CM DX | E08.x-E13.x; G45.x- 46.x; | Cerebrovascular |
| | 60.x-I79.x; I96; Z9582.x | disease |
| ICD-9-PROC | 3848 | Cerebrovascular |
| 7 | | disease |
| ICD-10-PROC | 04R.x-04RY4KZ | Cerebrovascular |
| | | disease |
| ICD-9-CM DX | 338.x | Chronic pain |
| ICD-10-CM DX | G89.x | Chronic pain |
| ICD-9-CM DX | 428.x | Congestive heart failure |
| ICD-10-CM DX | I09.x-I13.x; I50.x; R57.x | Congestive heart failure |
| ICD-9-CM DX | 49.x; 5064; 51.x; 7702 | COPD/asthma |
| ICD-10-CM DX | J4.x- J479 | COPD/asthma |
| ICD-9-CM DX | 410.x-4149; 433.x | Coronary artery/heart disease |
| ICD-10-CM DX | I20.x-I259; 63.x-I6529; Z955; Z9861 | Coronary artery/heart disease |
| ICD-10-CM DX | 250.x | Diabetes |
| ICD-9-CM DX | E10.x; E11.x; E13.x | Diabetes |
| ICD-10-CM DX | 345.x | Epilepsy |
| ICD-9-CM DX | G40.x-G40B19 | Epilepsy |
| ICD-10-CM DX | 00.x-129; 2515; 271.x-2892; 3064; 4474; | GI disorders |
| ICD-9-CWI DX | 45.x; 53.x-57.x; 61.x; 75.x; 78.x; 893.x; | Of disorders |
| | 997.x | |
| ICD-10-CM DX | A0.x; A2.x; A4.x; A5.x; B0x; B3.x; B6.x; | GI disorders |
| ICD-10-CWI DX | B7.x-B8.x; E164; E73.x-E74.x; I85.x- | GI disorders |
| | 1880; K2.x-K6.x; K9.x; N8.x; Q3.x-Q4.x; | |
| | Q7.x; R10.x-R198 | |
| ICD-9-CM DX | V08, 042, 07953 | HIV |
| ICD-10-CM DX | Z21, B20, B9735 | HIV |
| ICD-9-CM DX | 401.x-404.93 | Hypertension |
| ICD-10-CM DX | I10.x-I132 | Hypertension |
| ICD-9-CM DX | 346.x | Migraine |
| ICD-10-CM DX | G430.x-G324B1 | Migraine |
| ICD-9-CM DX | 278.0x | Obesity |
| ICD-10-CM DX | E66.x | Obesity |
| ICD-10-CM DX | 715.x; 7330.x | Osteoarthritis/osteoporosis |
| ICD-10-CM DX | M15.x-M19.x; M800.x; M81.x | Osteoarthritis/osteoporosis |
| ICD-9-CM DX | 331.82-33.2x | Parkinson's disease |
| ICD-9-CM DX | G20.x-G3183 | Parkinson's disease |
| ICD-10-CM DX | | Thyroid disease |
| | 240.x-2469 | , |
| ICD-10-CM DX | E00.x-E079 | Thyroid disease |

## Appendix 4: OPTION-12 Questionnaire

| 1 | The clinician draws attention to an identified problem as | Yes | No |
|---|---|---|---|
| | one that requires a decision making process. | 1 | 0 |
| 2 | The clinician states that there is more than one way to deal | Yes | No |
| | with the identified problem ('equipoise'). | 1 | 0 |
| 3 | The clinician assesses the patient's preferred approach to | Yes | No<br>0 |
| | receiving information to assist decision making (e.g. discussion, reading printed material, assessing graphical | ' | U |
| | data, using videotapes or other media). | | |
| 4 | The clinician <i>lists</i> 'options', which can include the choice of | Yes | No |
| | 'no action'. | 1 | 0 |
| 5 | The clinician explains the pros and cons of options to the | Yes | No |
| _ | patient (taking 'no action' is an option). | 1 | 0 |
| 6 | The clinician explores the patient's expectations (or ideas) | Yes | No<br>0 |
| | about how the problem(s) are to be managed. | ' | Ů |
| 7 | The clinician explores the patient's concerns (fears) about | Yes | No |
| | how problem(s) are to be managed. | 1 | 0 |
| 8 | The clinician checks that the patient has understood the | Yes | No |
| | information. | 1 | 0 |
| 9 | The clinician offers the patient explicit opportunities to ask | Yes | No |
| | questions during the decision making process. | 1 | 0 |
| 10 | The clinician elicits the patient's preferred level of | Yes | No |
| | involvement in decision-making. | 1 | 0 |
| 11 | The clinician indicates the need for a decision making (or | Yes | No |
| | deferring) stage. | 1 | 0 |
| 12 | The clinician indicates the need to review the decision (or | Yes | No |
| | deferment). | 1 | 0 |